CLINICAL TRIAL: NCT00972725
Title: A Study to Evaluate the Safety and Immunogenicity of a Booster Dose of GSK Biologicals' HIV Candidate Vaccine (732461) After Administration of Chloroquine in Healthy Adults.
Brief Title: Evaluation of the Immune Response of a HIV Candidate Vaccine After Administration of One Chloroquine Dose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113165
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-03

CONDITIONS: AIDS
Keywords: Chloroquine; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Chloroquine

ARMS (2):
- GSK732461+Nivaquine Group (Experimental): Subjects received a single dose of Nivaquine® tablets orally, 2 days prior to receiving a booster dose of the GSK732461 vaccine.
  Interventions: Biological: GSK Biologicals' HIV vaccine (732461); Drug: Chloroquine
- GSK732461 Group (Active Comparator): Subjects received a booster dose of the GSK732461 vaccine intramuscularly, in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' HIV vaccine (732461)

INTERVENTIONS:
Biological: GSK Biologicals' HIV vaccine (732461) — 1 dose intramuscular injection
Drug: Chloroquine — One dose of 300 mg
  Other Names: Nivaquine®
  Arms: GSK732461+Nivaquine Group

SUMMARY:
The purpose of this study is to evaluate the safety and reactogenicity of one booster dose of a HIV candidate vaccine after administration of one oral dose of chloroquine.

DETAILED DESCRIPTION:
The Protocol Posting has been updated following Protocol amendment 1, October 2009.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 18 to 52 years of age at the time of vaccination.
* Written informed consent prior to any study related procedure on the subject.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Good general health without significant medical history or physical examination findings.
* Negative for anti-HBc and anti-Hepatitis C Virus antibodies.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception until study completion.
* Previous participation and completion of the study NCT00434512.
* Cellular and humoral immune responder to vaccines administered in study NCT00434512.
* Subjects must be willing to accept HIV test results. Individuals who elect not to receive test results will not be enrolled.

Exclusion Criteria:

* Clinically significant laboratory value above normal range for blood urea nitrogen, creatinine, alanine aminotransferase and aspartate aminotransferase, or clinically significant laboratory value above or below normal range for Hemoglobin, as per investigator judgment.
* Women who are pregnant or breast-feeding.
* Receipt of live attenuated vaccines within 30 days of vaccination.
* Receipt of medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) or allergy treatment with antigen injections (including a tuberculin skin test) within <= 21days preceding and planned <= 21 days following the study vaccine administration.
* Receipt of blood products 120 days prior to vaccination.
* Receipt of immunoglobulin 120 days prior to vaccination.
* Subject has donated blood in the last 3 months.
* Bleeding disorder that was diagnosed by a physician; e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first.
* History of serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema and abdominal pain.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/product.
* History of serious allergic reaction to any substance requiring hospitalization or emergency medical care.
* History of hypersensitivity against chloroquine or any components of the drug.
* History of hypersensitivity against aminoglycosides.
* Ophthalmologic findings at screening.
* Previous administration of 4-aminoquinoline in the previous year or for a duration of more than 1 year.
* History of Glucose-6-Phosphate Dehydrogenase deficiency.
* History of hematopoietic disease.
* History of Myasthenia gravis.
* History of any serious neurological disorder or seizure.
* History of immunodeficiency or immune-mediated disorders, including active psoriasis.
* History of type I or type II diabetes mellitus including cases controlled with diet alone.
* Thyroid disease including history of thyroidectomy and diagnoses requiring medication.
* Asthma requiring daily steroid or long acting β-agonist prevention.
* Unstable asthma defined as:
* Sudden acute attacks occurring in less than three hours without an obvious trigger.
* Hospitalization for asthma in the last two years.
* Food- or wine-induced asthma.
* Known sensitivity to sulfites or aspirin.
* History of major congenital defect.
* History of chronic fatigue syndrome or fibromyalgia.
* History of malignancy.
* Splenectomy.
* Morbid obesity.
* Clinically relevant hypertension.
* Subjects with a history of, or current, alcohol or substance abuse.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous inclusion in a HIV vaccines trial other than study NCT00434512.
* Subject is seropositive for HIV, as determined by the test results performed.

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12-01; Primary Completion 2010-10-04 (Actual); Study Completion 2010-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels G, Bourguignon P, Willekens J, Janssens M, Clement F, Didierlaurent AM, Fissette L, Roman F, Boutriau D. Immunogenicity and safety of a booster dose of an investigational adjuvanted polyprotein HIV-1 vaccine in healthy adults and effect of administration of chloroquine. Clin Vaccine Immunol. 2014 Mar;21(3):302-11. doi: 10.1128/CVI.00617-13. Epub 2014 Jan 3. PMID 24391139

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of all the subjects planned for enrollment, only 28 were included in the analyses and hence started the study.
Period: Overall Study
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.1 (5.33) | 24.3 (3.73) | 24.67 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Frequency of Cluster of Differentiation 8 (CD8+) T Cells Expressing at Least One Cytokine to at Least 1, 2, 3 or All 4 Antigens
Description: Among expressed cytokines were interleukin-2 (IL-2), tumour necrosis factor alpha (TNF-α) and interferon gamma (INF-γ), as determined by intracellular cytokine staining (ICS).
Time Frame: At Day 14
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 13
Participants
  At least 1 antigen, Day 14 | 1 | 3
  At least 2 antigens, Day 14 | 0 | 0
  At least 3 antigens, Day 14 | 0 | 0
  At least 4 antigens, Day 14 | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7 Day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  Any Pain | 13 | 14
  Grade 3 Pain | 1 | 2
  Any Redness | 3 | 6
  Grade 3 Redness | 0 | 1
  Any Swelling | 3 | 5
  Grade 3 Swelling | 0 | 2

3. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain] and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7 Day (Days 0-6) post-vaccination period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  Any Fatigue | 9 | 14
  Grade 3 Fatigue | 3 | 3
  Related Fatigue | 9 | 11
  Any Gastrointestinal | 6 | 5
  Grade 3 Gastrointestinal | 1 | 0
  Related Gastrointestinal | 4 | 3
  Any Headache | 9 | 13
  Grade 3 Headache | 3 | 0
  Related Headache | 8 | 10
  Any Temperature | 8 | 10
  Grade 3 Temperature | 0 | 1
  Related Temperature | 7 | 9

4. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 32 Day (Days 2-29) post-chloroquine administration and during the 30 Day (Days 0-29) post-vaccine administration period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  Any AEs | 8 | 13
  Grade 3 AEs | 3 | 2
  Related AEs | 5 | 8

5. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 360)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants | 0 | 0

6. Primary Outcome: Number of Subjects With AEs of Specific Interest and Immune-Mediated Disorders (IMDs)
Description: Adverse events of specific interest include auto-immune diseases (AID) and immune mediated disorders such as neurological/demyelinating events, rheumatic and connective diseases, autoimmune endocrine diseases, inflammatory bowel diseases, autoimmune blood disorders, inflammatory skin disorders, other autoimmune/inflammatory events.
Time Frame: During the entire study period (from Day 0 up to Day 360)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants | 0 | 0

7. Primary Outcome: Levels of Haematological and Biochemical Parameters
Description: Among haematological and biochemical parameters determined were alanine aminotransferase [ALT], aspartate aminotransferase [ASA], basophils [BASO], creatinine [CREA], eosinophils [EOS], haematocrit [HAEM], haemoglobin [HAEMO], lymphocytes [LYMPH], monocytes [MONO], neutrophils [NEU], platelets [PLA], red blood cells [RBC], urea [UR] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed in relation to normal laboratory values were - unknown, below, within and above.
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  ALT, Unknown | 0 | 0
  ALT, Below | 0 | 0
  ALT, Within | 13 | 15
  ALT, Above | 0 | 0
  ASA, Unknown | 0 | 0
  ASA, Below | 0 | 0
  ASA, Within | 13 | 15
  ASA, Above | 0 | 0
  BASO, Unknown | 0 | 0
  BASO, Below | 3 | 4
  BASO, Within | 10 | 11
  BASO, Above | 0 | 0
  CREA, Unknown | 0 | 0
  CREA, Below | 0 | 0
  CREA, Within | 12 | 14
  CREA, Above | 1 | 1
  EOS, Unknown | 0 | 0
  EOS, Below | 1 | 1
  EOS, Within | 12 | 14
  EOS, Above | 0 | 0
  HAEM, Unknown | 0 | 0
  HAEM, Below | 1 | 0
  HAEM, Within | 12 | 15
  HAEM, Above | 0 | 0
  HAEMO, Unknown | 0 | 0
  HAEMO, Below | 0 | 0
  HAEMO, Within | 12 | 15
  HAEMO, Above | 1 | 0
  LYMPH, Unknown | 0 | 0
  LYMPH, Below | 1 | 3
  LYMPH, Within | 12 | 12
  LYMPH, Above | 0 | 0
  MONO, Unknown | 0 | 0
  MONO, Below | 0 | 0
  MONO, Within | 13 | 14
  MONO, Above | 0 | 1
  NEU, Unknown | 0 | 0
  NEU, Below | 2 | 0
  NEU, Within | 11 | 13
  NEU, Above | 0 | 2
  PLA, Unknown | 0 | 0
  PLA, Below | 0 | 0
  PLA, Within | 13 | 14
  PLA, Above | 0 | 1
  RBC, Unknown | 0 | 0
  RBC, Below | 0 | 0
  RBC, Within | 13 | 15
  RBC, Above | 0 | 0
  UR, Unknown | 0 | 0
  UR, Below | 0 | 0
  UR, Within | 13 | 15
  UR, Above | 0 | 0
  WBC, Unknown | 0 | 0
  WBC, Below | 0 | 0
  WBC, Within | 13 | 13
  WBC, Above | 0 | 2

8. Primary Outcome: Levels of Haematological and Biochemical Parameters
Description: as for outcome 7
Time Frame: At Day 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  ALT, Unknown | 0 | 0
  ALT, Below | 0 | 0
  ALT, Within | 13 | 15
  ALT, Above | 0 | 0
  ASA, Unknown | 0 | 0
  ASA, Below | 0 | 0
  ASA, Within | 13 | 15
  ASA, Above | 0 | 0
  BASO, Unknown | 0 | 0
  BASO, Below | 3 | 1
  BASO, Within | 10 | 14
  BASO, Above | 0 | 0
  CREA, Unknown | 0 | 0
  CREA, Below | 1 | 1
  CREA, Within | 11 | 12
  CREA, Above | 1 | 2
  EOS, Unknown | 1 | 1
  EOS, Below | 1 | 1
  EOS, Within | 0 | 0
  EOS, Above | 1 | 0
  HAEM, Unknown | 0 | 0
  HAEM, Below | 0 | 0
  HAEM, Within | 13 | 15
  HAEM, Above | 0 | 0
  HAEMO, Unknown | 0 | 0
  HAEMO, Below | 0 | 0
  HAEMO, Within | 13 | 15
  HAEMO, Above | 0 | 0
  LYMPH, Unknown | 0 | 0
  LYMPH, Below | 0 | 0
  LYMPH, Within | 13 | 15
  LYMPH, Above | 0 | 0
  MONO, Unknown | 0 | 0
  MONO, Below | 0 | 0
  MONO, Within | 11 | 15
  MONO, Above | 2 | 0
  NEU, Unknown | 0 | 0
  NEU, Below | 2 | 1
  NEU, Within | 10 | 14
  NEU, Above | 1 | 0
  PLA, Unknown | 0 | 0
  PLA, Below | 0 | 0
  PLA, Within | 13 | 14
  PLA, Above | 0 | 1
  RBC, Unknown | 0 | 0
  RBC, Below | 0 | 0
  RBC, Within | 13 | 15
  RBC, Above | 0 | 0
  UR, Unknown | 0 | 0
  UR, Below | 0 | 0
  UR, Within | 12 | 15
  UR, Above | 1 | 0
  WBC, Unknown | 0 | 0
  WBC, Below | 0 | 0
  WBC, Within | 12 | 15
  WBC, Above | 1 | 0

9. Primary Outcome: Levels of Haematological and Biochemical Parameters
Description: as for outcome 7
Time Frame: At Day 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  ALT, Unknown | 0 | 0
  ALT, Below | 0 | 0
  ALT, Within | 13 | 15
  ALT, Above | 0 | 0
  ASA, Unknown | 0 | 0
  ASA, Below | 0 | 0
  ASA, Within | 12 | 15
  ASA, Above | 1 | 0
  BASO, Unknown | 1 | 0
  BASO, Below | 2 | 2
  BASO, Within | 9 | 12
  BASO, Above | 1 | 1
  CREA, Unknown | 0 | 0
  CREA, Below | 0 | 0
  CREA, Within | 13 | 15
  CREA, Above | 0 | 0
  EOS, Unknown | 1 | 0
  EOS, Below | 0 | 0
  EOS, Within | 11 | 15
  EOS, Above | 1 | 0
  HAEM, Unknown | 1 | 0
  HAEM, Below | 0 | 0
  HAEM, Within | 12 | 15
  HAEM, Above | 0 | 0
  HAEMO, Unknown | 1 | 0
  HAEMO, Below | 0 | 0
  HAEMO, Within | 12 | 15
  HAEMO, Above | 0 | 0
  LYMPH, Unknown | 1 | 0
  LYMPH, Below | 1 | 1
  LYMPH, Within | 11 | 14
  LYMPH, Above | 0 | 0
  MONO, Unknown | 1 | 0
  MONO, Below | 0 | 0
  MONO, Within | 12 | 14
  MONO, Above | 0 | 1
  NEU, Unknown | 1 | 0
  NEU, Below | 3 | 0
  NEU, Within | 9 | 15
  NEU, Above | 0 | 0
  PLA, Unknown | 1 | 0
  PLA, Below | 0 | 0
  PLA, Within | 12 | 14
  PLA, Above | 0 | 1
  RBC, Unknown | 1 | 0
  RBC, Below | 0 | 0
  RBC, Within | 12 | 15
  RBC, Above | 0 | 0
  UR, Unknown | 0 | 0
  UR, Below | 1 | 0
  UR, Within | 12 | 15
  UR, Above | 0 | 0
  WBC, Unknown | 1 | 0
  WBC, Below | 1 | 0
  WBC, Within | 11 | 15
  WBC, Above | 0 | 0

10. Primary Outcome: Levels of Haematological and Biochemical Parameters
Description: as for outcome 7
Time Frame: At Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 15
Participants
  ALT, Unknown | 0 | 0
  ALT, Below | 0 | 0
  ALT, Within | 13 | 15
  ALT, Above | 0 | 0
  ASA, Unknown | 0 | 0
  ASA, Below | 0 | 0
  ASA, Within | 13 | 15
  ASA, Above | 0 | 0
  BASO, Unknown | 0 | 0
  BASO, Below | 1 | 2
  BASO, Within | 12 | 13
  BASO, Above | 0 | 0
  CREA, Unknown | 0 | 0
  CREA, Below | 0 | 0
  CREA, Within | 13 | 15
  CREA, Above | 0 | 0
  EOS, Unknown | 0 | 0
  EOS, Below | 1 | 0
  EOS, Within | 11 | 14
  EOS, Above | 1 | 1
  HAEM, Unknown | 0 | 0
  HAEM, Below | 0 | 0
  HAEM, Within | 13 | 15
  HAEM, Above | 0 | 0
  HAEMO, Unknown | 0 | 0
  HAEMO, Below | 0 | 0
  HAEMO, Within | 13 | 15
  HAEMO, Above | 0 | 0
  LYMPH, Unknown | 0 | 0
  LYMPH, Below | 1 | 3
  LYMPH, Within | 11 | 12
  LYMPH, Above | 1 | 0
  MONO, Unknown | 0 | 0
  MONO, Below | 0 | 0
  MONO, Within | 13 | 14
  MONO, Above | 0 | 1
  NEU, Unknown | 0 | 0
  NEU, Below | 2 | 1
  NEU, Within | 10 | 14
  NEU, Above | 1 | 0
  PLA, Unknown | 0 | 0
  PLA, Below | 0 | 0
  PLA, Within | 13 | 14
  PLA, Above | 0 | 1
  RBC, Unknown | 0 | 0
  RBC, Below | 0 | 0
  RBC, Within | 13 | 15
  RBC, Above | 0 | 0
  UR, Unknown | 0 | 0
  UR, Below | 0 | 0
  UR, Within | 13 | 15
  UR, Above | 0 | 0
  WBC, Unknown | 0 | 0
  WBC, Below | 0 | 0
  WBC, Within | 12 | 15
  WBC, Above | 1 | 0

11. Secondary Outcome: Magnitude of Antigen Specific CD8+ T Cells Expressing at Least One Cytokine
Description: Magnitude was defined as the frequency of CD8+ T cells group-specific antigen (Gag) proteins 17, 24; negative regulatory factor (Nef); reverse transcriptase (RT) and fusion protein of all 4 antigens (F4co). Determination of F4co was done by stimulating the F4 antigen with a peptide pool spanning (pool_F4co) or by adding individual frequencies of the CD8+ T cell response to each of the 4 antigens (F4co_est). Among the cytokines expressed were IL-2, TNF-α and INF-γ.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, D0 | 79.00 [54.00 to 140.00] | 89.00 [40.00 to 225.00]
  RT, D7: number analyzed (Participants) | 12 | 13
  RT, D7 | 127.50 [49.00 to 227.00] | 137.00 [70.00 to 168.00]
  RT, D14: number analyzed (Participants) | 13 | 13
  RT, D14 | 94.00 [53.00 to 214.00] | 102.00 [40.00 to 187.00]
  RT, D30: number analyzed (Participants) | 11 | 13
  RT, D30 | 57.00 [48.00 to 117.00] | 85.00 [14.00 to 113.00]
  RT, D180 | 14.00 [14.00 to 44.00] | 48.50 [33.00 to 71.00]
  Nef, D0 | 75.00 [46.00 to 121.00] | 71.00 [36.00 to 152.00]
  Nef, D7: number analyzed (Participants) | 12 | 13
  Nef, D7 | 63.50 [30.00 to 146.00] | 84.00 [44.00 to 130.00]
  Nef, D14: number analyzed (Participants) | 13 | 13
  Nef, D14 | 123.00 [93.00 to 184.00] | 99.00 [65.00 to 117.00]
  Nef, D30: number analyzed (Participants) | 11 | 13
  Nef, D30 | 61.00 [38.00 to 116.00] | 116.00 [74.00 to 146.00]
  Nef, D180 | 39.00 [14.00 to 74.00] | 66.00 [49.00 to 166.00]
  P17, D0 | 104.00 [41.00 to 127.00] | 76.00 [33.00 to 165.00]
  P17, D7: number analyzed (Participants) | 12 | 13
  P17, D7 | 109.50 [52.50 to 136.50] | 88.00 [42.00 to 113.00]
  P17, D14: number analyzed (Participants) | 13 | 13
  P17, D14 | 124.00 [38.00 to 178.00] | 84.00 [52.00 to 169.00]
  P17, D30: number analyzed (Participants) | 11 | 13
  P17, D30 | 18.00 [14.00 to 72.00] | 98.00 [49.00 to 120.00]
  P17, D180 | 55.00 [18.00 to 91.00] | 80.00 [68.00 to 142.00]
  P24, D0 | 68.00 [44.00 to 96.00] | 77.50 [14.00 to 126.00]
  P24, D7: number analyzed (Participants) | 12 | 13
  P24, D7 | 93.50 [21.50 to 159.50] | 54.00 [40.00 to 94.00]
  P24, D14: number analyzed (Participants) | 13 | 13
  P24, D14 | 83.00 [68.00 to 105.00] | 91.00 [49.00 to 106.00]
  P24, D30: number analyzed (Participants) | 11 | 13
  P24, D30 | 120.00 [73.00 to 134.00] | 81.00 [44.00 to 119.00]
  P24, D180 | 62.00 [14.00 to 102.00] | 45.00 [14.00 to 79.00]
  Pool_F4co, D0 | 76.00 [36.00 to 120.00] | 148.00 [73.00 to 201.00]
  Pool_F4co, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, D7 | 218.50 [81.50 to 242.50] | 129.00 [58.00 to 158.00]
  Pool_F4co, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, D14 | 92.00 [55.00 to 129.00] | 118.00 [76.00 to 168.00]
  Pool_F4co, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, D30 | 68.00 [16.00 to 132.00] | 122.00 [81.00 to 144.00]
  Pool_F4co, D180 | 65.00 [14.00 to 156.00] | 74.00 [50.00 to 98.00]
  F4co_est, D0 | 373.00 [271.00 to 453.00] | 398.00 [224.00 to 552.00]
  F4co_est, D7: number analyzed (Participants) | 12 | 13
  F4co_est, D7 | 448.50 [240.00 to 619.00] | 451.00 [329.00 to 534.00]
  F4co_est, D14: number analyzed (Participants) | 13 | 13
  F4co_est, D14 | 478.00 [313.00 to 554.00] | 450.00 [338.00 to 539.00]
  F4co_est, D30: number analyzed (Participants) | 11 | 13
  F4co_est, D30 | 290.00 [246.00 to 429.00] | 380.00 [241.00 to 555.00]
  F4co_est, D180 | 226.00 [108.00 to 299.00] | 287.50 [230.00 to 374.00]

12. Secondary Outcome: Frequency of Antigen (RT) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: Cytokine/marker co-expression profile was defined as the antigen-specific CD8+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or cluster of differentiation 40-ligand (CD40-L) cytokines as determined by ICS.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, CD40L+, D0 | 146.00 [42.00 to 228.00] | 123.00 [1.00 to 179.00]
  RT, CD40L+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+, D7 | 121.50 [1.00 to 272.00] | 168.00 [89.00 to 389.00]
  RT, CD40L+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+, D14 | 91.00 [11.00 to 177.00] | 1.00 [1.00 to 83.00]
  RT, CD40L+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+, D30 | 113.00 [1.00 to 238.00] | 27.00 [1.00 to 190.00]
  RT, CD40L+, D180 | 1.00 [1.00 to 100.00] | 52.50 [1.00 to 178.00]
  RT, IL2+, D0 | 31.00 [1.00 to 42.00] | 1.00 [1.00 to 79.00]
  RT, IL2+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+, D7 | 32.50 [1.00 to 55.00] | 1.00 [1.00 to 71.00]
  RT, IL2+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+, D14 | 64.00 [1.00 to 87.00] | 32.00 [1.00 to 60.00]
  RT, IL2+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+, D30 | 3.00 [1.00 to 54.00] | 1.00 [1.00 to 36.00]
  RT, IL2+, D180 | 1.00 [1.00 to 27.00] | 1.00 [1.00 to 31.00]
  RT, TNF+, D0 | 1.00 [1.00 to 28.00] | 1.00 [1.00 to 1.00]
  RT, TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, TNF+, D7 | 1.00 [1.00 to 19.50] | 34.00 [1.00 to 82.00]
  RT, TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, TNF+, D14 | 1.00 [1.00 to 21.00] | 1.00 [1.00 to 30.00]
  RT, TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, TNF+, D30 | 1.00 [1.00 to 30.00] | 1.00 [1.00 to 7.00]
  RT, TNF+, D180, | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IFN+, D0 | 1.00 [1.00 to 43.00] | 1.00 [1.00 to 40.00]
  RT, IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IFN+, D7 | 1.00 [1.00 to 31.00] | 1.00 [1.00 to 34.00]
  RT, IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IFN+, D14 | 14.00 [1.00 to 30.00] | 1.00 [1.00 to 1.00]
  RT, IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IFN+, D30 | 4.00 [1.00 to 30.00] | 1.00 [1.00 to 1.00]
  RT, IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 20.00]
  RT, CD40L+IL2+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

13. Secondary Outcome: Frequency of Antigen (RT) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: Cytokine/marker co-expression profile was defined as the antigen-specific CD8+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L cytokines as determined by ICS.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 20.00]
  RT, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, TNF+IFN+, D7 | 1.00 [1.00 to 31.50] | 1.00 [1.00 to 20.00]
  RT, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 37.00]
  RT, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+TNF+IFN+, D7 | 1.00 [1.00 to 6.50] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

14. Secondary Outcome: Frequency of Antigen (Nef) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 12
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Nef, CD40L+, D0 | 155.00 [45.00 to 226.00] | 72.50 [1.00 to 166.00]
  Nef, CD40L+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+, D7 | 90.50 [33.50 to 157.00] | 173.00 [30.00 to 280.00]
  Nef, CD40L+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+, D14 | 122.00 [82.00 to 231.00] | 10.00 [1.00 to 81.00]
  Nef, CD40L+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+, D30 | 191.00 [1.00 to 373.00] | 30.00 [1.00 to 107.00]
  Nef, CD40L+, D180 | 134.00 [45.00 to 174.00] | 43.50 [1.00 to 169.00]
  Nef, IL2+, D0 | 1.00 [1.00 to 55.00] | 9.50 [1.00 to 70.00]
  Nef, IL2+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+, D7 | 22.00 [1.00 to 43.50] | 1.00 [1.00 to 30.00]
  Nef, IL2+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+, D14 | 40.00 [1.00 to 78.00] | 59.00 [1.00 to 74.00]
  Nef, IL2+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+, D30 | 1.00 [1.00 to 21.00] | 1.00 [1.00 to 74.00]
  Nef, IL2+, D180 | 1.00 [1.00 to 1.00] | 26.50 [1.00 to 100.00]
  Nef, TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 6.00]
  Nef, TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, TNF+, D7 | 1.00 [1.00 to 29.50] | 4.00 [1.00 to 60.00]
  Nef, TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, TNF+, D14 | 1.00 [1.00 to 35.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, TNF+, D30 | 1.00 [1.00 to 39.00] | 1.00 [1.00 to 51.00]
  Nef, TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IFN+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 20.00]
  Nef, IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IFN+, D7 | 1.00 [1.00 to 34.00] | 1.00 [1.00 to 1.00]
  Nef, IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IFN+, D14 | 1.00 [1.00 to 26.00] | 1.00 [1.00 to 1.00]
  Nef, IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IFN+, D30 | 2.00 [1.00 to 31.00] | 1.00 [1.00 to 18.00]
  Nef, IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 36.00]
  Nef, CD40L+IL2+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  Nef, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 15.00]
  Nef, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

15. Secondary Outcome: Frequency of Antigen (Nef) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 13
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Nef, IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 35.00]
  Nef, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+TNF+, D30 | 1.00 [1.00 to 21.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

16. Secondary Outcome: Frequency of Antigen (p17) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 13
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P17, CD40L+, D0 | 65.00 [1.00 to 191.00] | 1.00 [1.00 to 158.00]
  P17, CD40L+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+, D7 | 40.50 [1.00 to 142.00] | 34.00 [1.00 to 128.00]
  P17, CD40L+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+, D14 | 1.00 [1.00 to 169.00] | 1.00 [1.00 to 33.00]
  P17, CD40L+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+, D30 | 7.00 [1.00 to 126.00] | 13.00 [1.00 to 165.00]
  P17, CD40L+, D180 | 44.00 [1.00 to 73.00] | 4.50 [1.00 to 50.00]
  P17, IL2+, D0 | 1.00 [1.00 to 28.00] | 1.00 [1.00 to 26.00]
  P17, IL2+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+, D7 | 7.50 [1.00 to 34.00] | 21.00 [1.00 to 34.00]
  P17, IL2+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+, D14 | 25.00 [1.00 to 92.00] | 33.00 [1.00 to 60.00]
  P17, IL2+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+, D30 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 35.00]
  P17, IL2+, D180 | 10.00 [1.00 to 61.00] | 39.00 [1.00 to 67.00]
  P17, TNF+, D0 | 1.00 [1.00 to 65.00] | 1.00 [1.00 to 7.00]
  P17, TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, TNF+, D7 | 1.00 [1.00 to 45.50] | 21.00 [1.00 to 68.00]
  P17, TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, TNF+, D14 | 1.00 [1.00 to 36.00] | 1.00 [1.00 to 2.00]
  P17, TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 50.00]
  P17, TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IFN+, D0 | 1.00 [1.00 to 31.00] | 1.00 [1.00 to 20.00]
  P17, IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IFN+, D7 | 1.00 [1.00 to 28.50] | 1.00 [1.00 to 1.00]
  P17, IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 20.00]
  P17, IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IFN+, D30 | 1.00 [1.00 to 22.00] | 1.00 [1.00 to 34.00]
  P17, IFN+, D180 | 3.00 [1.00 to 26.00] | 1.00 [1.00 to 23.00]
  P17, CD40L+IL2+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

17. Secondary Outcome: Frequency of Antigen (p17) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 13
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P17, IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 16.00]
  P17, IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, TNF+IFN+, D7 | 1.00 [1.00 to 7.50] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  p17, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

18. Secondary Outcome: Frequency of Antigen (p24) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 13
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P24, CD40L+, D0 | 178.00 [1.00 to 219.00] | 103.50 [1.00 to 163.00]
  P24, CD40L+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+, D7 | 61.50 [2.50 to 138.00] | 37.00 [1.00 to 219.00]
  P24, CD40L+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+, D14 | 100.00 [17.00 to 171.00] | 30.00 [1.00 to 130.00]
  P24, CD40L+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+, D30 | 1.00 [1.00 to 179.00] | 59.00 [1.00 to 133.00]
  P24, CD40L+, D180 | 16.00 [1.00 to 210.00] | 1.00 [1.00 to 37.00]
  P24, IL2+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 37.00]
  P24, IL2+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+, D7 | 7.50 [1.00 to 43.00] | 1.00 [1.00 to 26.00]
  P24, IL2+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+, D14 | 1.00 [1.00 to 54.00] | 1.00 [1.00 to 38.00]
  P24, IL2+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+, D30 | 1.00 [1.00 to 54.00] | 32.00 [1.00 to 73.00]
  P24, IL2+, D180 | 1.00 [1.00 to 53.00] | 1.00 [1.00 to 34.00]
  P24, TNF+, D0 | 1.00 [1.00 to 55.00] | 1.00 [1.00 to 1.00]
  P24, TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, TNF+, D7 | 1.00 [1.00 to 32.00] | 27.00 [1.00 to 55.00]
  P24, TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, TNF+, D14 | 1.00 [1.00 to 41.00] | 1.00 [1.00 to 1.00]
  P24, TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, TNF+, D30 | 1.00 [1.00 to 60.00] | 1.00 [1.00 to 23.00]
  P24, TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 21.00]
  P24, IFN+, D0 | 5.00 [1.00 to 55.00] | 1.00 [1.00 to 56.00]
  P24, IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IFN+, D7 | 1.00 [1.00 to 35.00] | 1.00 [1.00 to 1.00]
  P24, IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IFN+, D14 | 1.00 [1.00 to 36.00] | 1.00 [1.00 to 1.00]
  P24, IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IFN+, D30 | 25.00 [1.00 to 44.00] | 1.00 [1.00 to 42.00]
  P24, IFN+, D180 | 1.00 [1.00 to 25.00] | 1.00 [1.00 to 19.00]
  P24, CD40L+IL2+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

19. Secondary Outcome: Frequency of Antigen (p24) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 13
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P24, IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 34.00]
  P24, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

20. Secondary Outcome: Frequency of Antigen (pool_F4co) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: Cytokine/marker co-expression profile was defined as the antigen-specific CD8+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L cytokines as determined by ICS. Determination of F4co was done by stimulating the F4 antigen with a peptide pool spanning (pool_F4co) or by adding individual frequencies of the CD8+ T cell response to each of the 4 antigens (F4co_est).
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Pool_F4co, CD40L+, D0 | 114.00 [1.00 to 264.00] | 105.00 [1.00 to 256.00]
  Pool_F4co, CD40L+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+, D7 | 141.50 [37.50 to 235.00] | 185.00 [109.00 to 223.00]
  Pool_F4co, CD40L+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+, D14 | 113.00 [78.00 to 181.00] | 1.00 [1.00 to 69.00]
  Pool_F4co, CD40L+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+, D30 | 84.00 [7.00 to 251.00] | 69.00 [1.00 to 192.00]
  Pool_F4co, CD40L+, D180 | 61.00 [42.00 to 107.00] | 48.00 [1.00 to 173.00]
  Pool_F4co, IL2+, D0 | 1.00 [1.00 to 28.00] | 22.00 [1.00 to 54.00]
  Pool_F4co, IL2+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+, D7 | 26.00 [1.00 to 132.00] | 3.00 [1.00 to 85.00]
  Pool_F4co, IL2+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+, D14 | 31.00 [1.00 to 54.00] | 32.00 [15.00 to 84.00]
  Pool_F4co, IL2+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+, D30 | 1.00 [1.00 to 88.00] | 20.00 [1.00 to 68.00]
  Pool_F4co, IL2+, D180 | 27.00 [1.00 to 89.00] | 1.00 [1.00 to 57.00]
  Pool_F4co, TNF+, D0 ] | 1.00 [1.00 to 32.00] | 1.00 [1.00 to 23.00]
  Pool_F4co, TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, TNF+, D7 | 1.00 [1.00 to 28.50] | 5.00 [1.00 to 33.00]
  Pool_F4co, TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, TNF+, D14 | 2.00 [1.00 to 32.00] | 1.00 [1.00 to 72.00]
  Pool_F4co, TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, TNF+, D30 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 35.00]
  Pool_F4co, TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IFN+, D0 | 1.00 [1.00 to 17.00] | 28.00 [1.00 to 78.00]
  Pool_F4co, IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IFN+, D7 | 1.00 [1.00 to 15.00] | 14.00 [1.00 to 33.00]
  Pool_F4co, IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IFN+, D14 | 5.00 [1.00 to 33.00] | 1.00 [1.00 to 27.00]
  Pool_F4co, IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IFN+, D30 | 1.00 [1.00 to 1.00] | 17.00 [1.00 to 38.00]
  Pool_F4co, IFN+, D180 | 1.00 [1.00 to 41.00] | 1.00 [1.00 to 33.00]
  Pool_F4co, CD40L+IL2+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+, D7 | 1.00 [1.00 to 31.50] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IFN+, D7 | 1.00 [1.00 to 27.50] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

21. Secondary Outcome: Frequency of Antigen (pool_F4co) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 20
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Pool_F4co, IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+TNF+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+TNF+, D14 | 1.00 [1.00 to 28.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, TNF+IFN+, D0 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, TNF+IFN+, D7 | 1.00 [1.00 to 13.00] | 1.00 [1.00 to 14.00]
  Pool_F4co, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 23.00]
  Pool_F4co, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+TNF+, D7 | 1.00 [1.00 to 7.50] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+TNF+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+TNF+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+TNF+IFN+, D180 [ | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

22. Secondary Outcome: Frequency of Antigen (F4co_est) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 20
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  F4co_est, CD40L+, D0 | 608.00 [206.00 to 746.00] | 301.00 [139.00 to 603.00]
  F4co_est, CD40L+, D7 | 359.50 [238.00 to 603.50] | 532.00 [191.00 to 834.00]
  F4co_est, CD40L+, D14 | 375.00 [237.00 to 717.00] | 201.00 [94.00 to 305.00]
  F4co_est, CD40L+, D30 | 347.00 [21.00 to 783.00] | 242.00 [71.00 to 693.00]
  F4co_est, CD40L+, D180 | 278.00 [100.00 to 534.00] | 150.00 [67.00 to 346.00]
  F4co_est, IL2+, D0 | 77.00 [45.00 to 131.00] | 64.00 [26.00 to 143.00]
  F4co_est, IL2+, D7 | 129.00 [41.00 to 164.00] | 84.00 [35.00 to 188.00]
  F4co_est, IL2+, D14 | 122.00 [68.00 to 305.00] | 141.00 [71.00 to 253.00]
  F4co_est, IL2+, D30 | 22.00 [4.00 to 151.00] | 73.00 [38.00 to 168.00]
  F4co_est, IL2+, D180 | 85.00 [6.00 to 128.00] | 127.50 [46.00 to 169.00]
  F4co_est, TNF+, D0 | 112.00 [4.00 to 163.00] | 9.50 [4.00 to 30.00]
  F4co_est, TNF+, D7 | 57.50 [17.00 to 140.00] | 176.00 [24.00 to 248.00]
  F4co_est, TNF+, D14 | 55.00 [4.00 to 147.00] | 4.00 [4.00 to 86.00]
  F4co_est, TNF+, D30 | 4.00 [4.00 to 160.00] | 67.00 [4.00 to 140.00]
  F4co_est, TNF+, D180 | 4.00 [4.00 to 28.00] | 14.50 [4.00 to 68.00]
  F4co_est, IFN+, D0 | 60.00 [8.00 to 105.00] | 58.50 [17.00 to 133.00]
  F4co_est, IFN+, D7 | 36.00 [4.00 to 133.50] | 29.00 [4.00 to 70.00]
  F4co_est, IFN+, D14 | 56.00 [39.00 to 86.00] | 21.00 [4.00 to 84.00]
  F4co_est, IFN+, D30 | 52.00 [8.00 to 130.00] | 22.00 [4.00 to 109.00]
  F4co_est, IFN+, D180 | 30.00 [6.00 to 66.00] | 23.50 [4.00 to 86.00]
  F4co_est, CD40L+IL2+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+, D7 | 4.00 [4.00 to 9.50] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+, D7 | 4.00 [4.00 to 36.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IFN+, D7 | 4.00 [4.00 to 23.50] | 5.00 [4.00 to 24.00]
  F4co_est, CD40L+IFN+, D14 | 4.00 [4.00 to 17.00] | 4.00 [4.00 to 30.00]
  F4co_est, CD40L+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IFN+, D180 | 4.00 [4.00 to 28.00] | 4.00 [4.00 to 22.00]

23. Secondary Outcome: Frequency of Antigen (F4co_est) Specific CD8+ T Cells Expressing at Least One Marker/ Cytokine
Description: as for outcome 20
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  F4co_est, IL2+TNF+, D0 | 4.00 [4.00 to 64.00] | 28.00 [4.00 to 43.00]
  F4co_est, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+TNF+, D7 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 23.00]
  F4co_est, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+TNF+, D14 | 4.00 [4.00 to 32.00] | 4.00 [4.00 to 23.00]
  F4co_est, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+TNF+, D30 | 4.00 [4.00 to 44.00] | 4.00 [4.00 to 27.00]
  F4co_est, IL2+TNF+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+IFN+, D7 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+IFN+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, TNF+IFN+, D0 | 4.00 [4.00 to 5.00] | 4.00 [4.00 to 43.00]
  F4co_est, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, TNF+IFN+, D7 | 15.50 [4.00 to 50.00] | 23.00 [4.00 to 40.00]
  F4co_est, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, TNF+IFN+, D14 | 4.00 [4.00 to 29.00] | 4.00 [4.00 to 29.00]
  F4co_est, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, TNF+IFN+, D30 | 4.00 [4.00 to 27.00] | 27.00 [4.00 to 78.00]
  F4co_est, TNF+IFN+, D180 | 4.00 [4.00 to 5.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+TNF+, D7 | 4.00 [4.00 to 25.50] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+TNF+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+TNF+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+IFN+, D7 | 4.00 [4.00 to 30.50] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+IFN+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+IFN+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+TNF+IFN+, D7 | 4.00 [4.00 to 9.50] | 4.00 [4.00 to 4.00]
  F4co_est, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40+TNF+IFN+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+TNF+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+TNF+IFN+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+TNF+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+TNF+IFN+, D7 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+TNF+IFN+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+TNF+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+TNF+IFN+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D7 | 4.00 [4.00 to 9.50] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D14 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D180 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]

24. Secondary Outcome: Number of Subjects With Frequency of Cluster of Differentiation (CD4+) T Cells Expressing at Least 2 Cytokines to at Least 1, 2, 3 or All 4 Antigens
Description: Among expressed cytokines were interleukin-2 (IL-2), tumour necrosis factor alpha (TNF-α) and interferon gamma (INF-γ), as determined by ICS.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
Participants
  1 antigen, Day 0 | 12 | 11
  1 antigen, Day 7: number analyzed (Participants) | 12 | 13
  1 antigen, Day 7 | 12 | 12
  1 antigen, Day 14: number analyzed (Participants) | 13 | 13
  1 antigen, Day 14 | 12 | 12
  1 antigen, Day 30: number analyzed (Participants) | 11 | 13
  1 antigen, Day 30 | 8 | 13
  1 antigen, Day 180 | 13 | 14
  2 antigens, Day 0 | 10 | 11
  2 antigens, Day 7: number analyzed (Participants) | 12 | 13
  2 antigens, Day 7 | 11 | 11
  2 antigens, Day 14: number analyzed (Participants) | 13 | 13
  2 antigens, Day 14 | 12 | 11
  2 antigens, Day 30: number analyzed (Participants) | 11 | 13
  2 antigens, Day 30 | 7 | 13
  2 antigens, Day 180 | 11 | 13
  3 antigens, Day 0 | 6 | 4
  3 antigens, Day 7: number analyzed (Participants) | 12 | 13
  3 antigens, Day 7 | 10 | 10
  3 antigens, Day 14: number analyzed (Participants) | 13 | 13
  3 antigens, Day 14 | 10 | 10
  3 antigens, Day 30: number analyzed (Participants) | 11 | 13
  3 antigens, Day 30 | 7 | 10
  3 antigens, Day 180 | 10 | 9
  4 antigens, Day 0 | 1 | 3
  4 antigens, Day 7: number analyzed (Participants) | 12 | 13
  4 antigens, Day 7 | 6 | 8
  4 antigens, Day 14: number analyzed (Participants) | 13 | 13
  4 antigens, Day 14 | 6 | 8
  4 antigens, Day 30: number analyzed (Participants) | 11 | 13
  4 antigens, Day 30 | 7 | 6
  4 antigens, Day 180 | 3 | 4

25. Secondary Outcome: Magnitude of Antigen Specific CD4+ T Cells Expressing at Least 2 Cytokines
Description: Magnitude was defined as the frequency of CD4+ T cells group-specific antigen (Gag) proteins 17, 24, negative regulatory factor (Nef), reverse transcriptase (RT) and fusion protein of all 4 antigens (F4co). Determination of F4co was done by stimulating the F4 antigen with a peptide pool spanning (pool_F4co) or by adding individual frequencies of the CD8+ T cell response to each of the 4 antigens (F4co_est). Among the cytokines expressed were IL-2, TNF-α and INF-γ.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, Day 0 | 846.00 [616.00 to 1252.00] | 1125.50 [373.00 to 2290.00]
  RT, Day 7: number analyzed (Participants) | 12 | 13
  RT, Day 7 | 2407.00 [1477.50 to 4566.00] | 3286.00 [1788.00 to 5334.00]
  RT, Day 14: number analyzed (Participants) | 13 | 13
  RT, Day 14 | 3162.00 [1393.00 to 4433.00] | 3461.00 [2931.00 to 3868.00]
  RT, Day 30: number analyzed (Participants) | 11 | 13
  RT, Day 30 | 2088.00 [54.00 to 4545.00] | 2459.00 [1897.00 to 3334.00]
  RT, Day 180 | 1205.00 [1037.00 to 2518.00] | 1684.00 [919.00 to 2566.00]
  Nef, Day 0 | 259.00 [206.00 to 310.00] | 161.00 [98.00 to 589.00]
  Nef, Day 7: number analyzed (Participants) | 12 | 13
  Nef, Day 7 | 586.50 [345.50 to 961.50] | 739.00 [324.00 to 1292.00]
  Nef, Day 14: number analyzed (Participants) | 13 | 13
  Nef, Day 14 | 890.00 [271.00 to 1362.00] | 560.00 [227.00 to 1223.00]
  Nef, Day 30: number analyzed (Participants) | 11 | 13
  Nef, Day 30 | 627.00 [84.00 to 1731.00] | 386.00 [199.00 to 945.00]
  Nef, Day 180 | 305.00 [245.00 to 518.00] | 306.50 [162.00 to 785.00]
  P17, Day 0 | 154.00 [121.00 to 264.00] | 176.00 [135.00 to 417.00]
  P17, Day 7: number analyzed (Participants) | 12 | 13
  P17, Day 7 | 464.00 [119.00 to 835.50] | 500.00 [127.00 to 1678.00]
  P17, Day 14: number analyzed (Participants) | 13 | 13
  P17, Day 14 | 453.00 [160.00 to 593.00] | 503.00 [200.00 to 1224.00]
  P17, Day 30: number analyzed (Participants) | 11 | 13
  P17, Day 30 | 397.00 [44.00 to 1207.00] | 346.00 [232.00 to 981.00]
  P17, Day 180 | 278.00 [123.00 to 423.00] | 523.00 [172.00 to 837.00]
  P24, Day 0 | 477.00 [322.00 to 642.00] | 434.00 [57.00 to 934.00]
  P24, Day 7: number analyzed (Participants) | 12 | 13
  P24, Day 7 | 872.50 [435.00 to 1700.00] | 911.00 [549.00 to 1507.00]
  P24, Day 14: number analyzed (Participants) | 13 | 13
  P24, Day 14 | 1198.00 [582.00 to 1653.00] | 827.00 [492.00 to 1569.00]
  P24, Day 30: number analyzed (Participants) | 11 | 13
  P24, Day 30 | 641.00 [152.00 to 1136.00] | 793.00 [492.00 to 1285.00]
  P24, Day 180 | 530.00 [396.00 to 714.00] | 536.50 [302.00 to 826.00]
  Pool_F4co, Day 0 | 1421.00 [965.00 to 2045.00] | 2006.50 [1135.00 to 4228.00]
  Pool_F4co, Day 7: number analyzed (Participants) | 12 | 13
  Pool_F4co, Day 7 | 3881.00 [2480.00 to 6982.00] | 5515.00 [4179.00 to 7947.00]
  Pool_F4co, Day 14: number analyzed (Participants) | 13 | 13
  Pool_F4co, Day 14 | 4898.00 [2446.00 to 7829.00] | 5651.00 [4961.00 to 6599.00]
  Pool_F4co, Day 30: number analyzed (Participants) | 11 | 13
  Pool_F4co, Day 30 | 3791.00 [322.00 to 6073.00] | 4138.00 [3485.00 to 5158.00]
  Pool_F4co, Day 180 | 2238.00 [1983.00 to 3956.00] | 2856.50 [2233.00 to 4441.00]
  F4co_est, Day 0 | 2000.00 [1492.00 to 2313.00] | 1974.50 [1195.00 to 4657.00]
  F4co_est, Day 7: number analyzed (Participants) | 12 | 13
  F4co_est, Day 7 | 4390.00 [2708.00 to 7841.00] | 6613.00 [4980.00 to 8883.00]
  F4co_est, Day 14: number analyzed (Participants) | 13 | 13
  F4co_est, Day 14 | 5272.00 [2772.00 to 8751.00] | 6035.00 [5437.00 to 7244.00]
  F4co_est, Day 30: number analyzed (Participants) | 11 | 13
  F4co_est, Day 30 | 4407.00 [354.00 to 7708.00] | 4589.00 [3458.00 to 5266.00]
  F4co_est, Day 180 | 2530.00 [2151.00 to 4596.00] | 3079.00 [2448.00 to 5123.00]

26. Secondary Outcome: Frequency of Antigen (RT) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: Cytokine/marker co-expression profile was defined as the antigen-specific CD4+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L cytokines as determined by ICS.
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, CD40L+, D0 | 163.00 [52.00 to 240.00] | 184.00 [13.00 to 299.00]
  RT, CD40L+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+, D7 | 1080.50 [603.00 to 2695.50] | 1209.00 [469.00 to 1534.00]
  RT, CD40L+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+, D14 | 522.00 [106.00 to 1170.00] | 748.00 [168.00 to 994.00]
  RT, CD40L+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+, D30 | 262.00 [1.00 to 869.00] | 309.00 [233.00 to 543.00]
  RT, CD40L+, D180 | 229.00 [159.00 to 346.00] | 249.00 [135.00 to 420.00]
  RT, IL2+, D0 | 1.00 [1.00 to 27.00] | 15.00 [12.00 to 82.00]
  RT, IL2+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+, D7 | 85.50 [58.00 to 130.50] | 42.00 [14.00 to 76.00]
  RT, IL2+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+, D14 | 97.00 [34.00 to 121.00] | 35.00 [15.00 to 80.00]
  RT, IL2+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+, D30 | 24.00 [1.00 to 69.00] | 36.00 [28.00 to 68.00]
  RT, IL2+, D180 | 41.00 [1.00 to 79.00] | 74.00 [41.00 to 104.00]
  RT, TNF+, D0 | 18.00 [1.00 to 143.00] | 61.50 [1.00 to 286.00]
  RT, TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, TNF+, D7 | 421.00 [130.50 to 504.50] | 312.00 [141.00 to 481.00]
  RT, TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, TNF+, D14 | 228.00 [149.00 to 264.00] | 318.00 [84.00 to 479.00]
  RT, TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, TNF+, D30 | 124.00 [2.00 to 191.00] | 231.00 [42.00 to 287.00]
  RT, TNF+, D180 | 74.00 [16.00 to 81.00] | 7.00 [1.00 to 54.00]
  RT, IFN+, D0 | 7.00 [1.00 to 24.00] | 13.00 [1.00 to 14.00]
  RT, IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IFN+, D7 | 91.50 [18.00 to 143.00] | 56.00 [13.00 to 81.00]
  RT, IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IFN+, D14 | 9.00 [1.00 to 16.00] | 16.00 [1.00 to 56.00]
  RT, IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IFN+, D30 | 1.00 [1.00 to 27.00] | 1.00 [1.00 to 14.00]
  RT, IFN+, D180 | 13.00 [1.00 to 53.00] | 12.50 [1.00 to 41.00]
  RT, CD40L+IL2+, D0 | 377.00 [149.00 to 579.00] | 315.00 [121.00 to 544.00]
  RT, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+, D7 | 924.00 [544.00 to 1793.50] | 1424.00 [549.00 to 2016.00]
  RT, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+, D14 | 922.00 [413.00 to 1702.00] | 990.00 [556.00 to 1286.00]
  RT, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+, D30 | 615.00 [1.00 to 1053.00] | 828.00 [516.00 to 1127.00]
  RT, CD40L+IL2+, D180 | 558.00 [447.00 to 866.00] | 797.50 [364.00 to 1013.00]
  RT, CD40L+TNF+, D0 | 41.00 [6.00 to 53.00] | 36.50 [14.00 to 110.00]
  RT, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+TNF+, D7 | 237.00 [103.00 to 469.00] | 315.00 [95.00 to 373.00]
  RT, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+TNF+, D14 | 300.00 [107.00 to 410.00] | 291.00 [199.00 to 432.00]
  RT, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+TNF+, D30 | 204.00 [36.00 to 314.00] | 137.00 [131.00 to 156.00]
  RT, CD40L+TNF+, D180 | 54.00 [21.00 to 68.00] | 40.50 [27.00 to 66.00]
  RT, CD40L+IFN+, D0 | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 1.00]
  RT, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IFN+, D7 | 69.00 [18.50 to 160.00] | 84.00 [14.00 to 126.00]
  RT, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IFN+, D14 | 27.00 [14.00 to 83.00] | 28.00 [14.00 to 69.00]
  RT, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IFN+, D30 | 14.00 [1.00 to 32.00] | 15.00 [14.00 to 30.00]
  RT, CD40L+IFN+, D180 | 1.00 [1.00 to 14.00] | 14.00 [1.00 to 24.00]

27. Secondary Outcome: Frequency of Antigen (RT) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  RT, IL2+TNF+, D0 | 14.00 [2.00 to 42.00] | 6.50 [1.00 to 43.00]
  RT, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+TNF+, D7 | 83.50 [45.00 to 159.00] | 37.00 [14.00 to 56.00]
  RT, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+TNF+, D14 | 53.00 [15.00 to 183.00] | 22.00 [1.00 to 103.00]
  RT, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+TNF+, D30 | 27.00 [1.00 to 48.00] | 55.00 [27.00 to 129.00]
  RT, IL2+TNF+, D180 | 26.00 [14.00 to 64.00] | 67.50 [41.00 to 94.00]
  RT, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+IFN+, D7 | 10.50 [1.00 to 14.50] | 1.00 [1.00 to 9.00]
  RT, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+IFN+, D14 | 1.00 [1.00 to 15.00] | 1.00 [1.00 to 14.00]
  RT, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  RT, IL2+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  RT, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  RT, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, TNF+IFN+, D7 | 18.00 [8.00 to 48.00] | 28.00 [1.00 to 37.00]
  RT, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, TNF+IFN+, D14 | 23.00 [1.00 to 41.00] | 14.00 [1.00 to 54.00]
  RT, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, TNF+IFN+, D30 | 14.00 [1.00 to 27.00] | 19.00 [9.00 to 29.00]
  RT, TNF+IFN+, D180 | 1.00 [1.00 to 14.00] | 15.00 [1.00 to 41.00]
  RT, CD40L+IL2+TNF+, D0 | 475.00 [218.00 to 664.00] | 474.50 [227.00 to 1308.00]
  RT, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+TNF+, D7 | 842.00 [588.50 to 1928.00] | 1575.00 [1013.00 to 2699.00]
  RT, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+TNF+, D14 | 1606.00 [707.00 to 2546.00] | 1901.00 [1551.00 to 2221.00]
  RT, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+TNF+, D30 | 1209.00 [19.00 to 2489.00] | 1297.00 [999.00 to 1791.00]
  RT, CD40L+IL2+TNF+, D180 | 471.00 [350.00 to 851.00] | 709.50 [485.00 to 1196.00]
  RT, CD40L+IL2+IFN+, D0 | 15.00 [1.00 to 55.00] | 12.50 [1.00 to 29.00]
  RT, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+IFN+, D7 | 89.50 [18.50 to 316.50] | 151.00 [56.00 to 169.00]
  RT, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+IFN+, D14 | 54.00 [25.00 to 113.00] | 84.00 [42.00 to 128.00]
  RT, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+IFN+, D30 | 30.00 [1.00 to 141.00] | 56.00 [15.00 to 102.00]
  RT, CD40L+IL2+IFN+, D180 | 68.00 [14.00 to 104.00] | 40.50 [26.00 to 78.00]
  RT, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 9.00] | 1.00 [1.00 to 14.00]
  RT, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+TNF+IFN+, D7 | 43.00 [27.50 to 86.00] | 56.00 [24.00 to 74.00]
  RT, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40+TNF+IFN+, D14 | 50.00 [30.00 to 81.00] | 28.00 [1.00 to 56.00]
  RT, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+TNF+IFN+, D30 | 27.00 [9.00 to 65.00] | 15.00 [14.00 to 42.00]
  RT, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 27.00]
  RT, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 12.00]
  RT, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, IL2+TNF+IFN+, D7 | 13.50 [1.00 to 25.00] | 14.00 [8.00 to 27.00]
  RT, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, IL2+TNF+IFN+, D14 | 8.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  RT, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 11.00] | 13.00 [1.00 to 14.00]
  RT, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 27.00] | 13.50 [1.00 to 27.00]
  RT, CD40L+IL2+TNF+IFN+, D0 | 57.00 [14.00 to 92.00] | 48.00 [1.00 to 151.00]
  RT, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  RT, CD40L+IL2+TNF+IFN+, D7 | 206.50 [72.50 to 600.50] | 213.00 [82.00 to 573.00]
  RT, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  RT, CD40L+IL2+TNF+IFN+, D14 | 254.00 [68.00 to 354.00] | 285.00 [152.00 to 393.00]
  RT, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  RT, CD40L+IL2+TNF+IFN+, D30 | 136.00 [1.00 to 499.00] | 237.00 [97.00 to 379.00]
  RT, CD40L+IL2+TNF+IFN+, D180 | 64.00 [52.00 to 236.00] | 87.50 [45.00 to 225.00]

28. Secondary Outcome: Frequency of Antigen (Nef) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Nef, CD40L+, D0 | 113.00 [1.00 to 311.00] | 1.00 [1.00 to 49.00]
  Nef, CD40L+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+, D7 | 339.00 [232.50 to 572.00] | 294.00 [94.00 to 402.00]
  Nef, CD40L+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+, D14 | 224.00 [109.00 to 557.00] | 219.00 [84.00 to 299.00]
  Nef, CD40L+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+, D30 | 193.00 [1.00 to 314.00] | 153.00 [14.00 to 245.00]
  Nef, CD40L+, D180 | 107.00 [52.00 to 173.00] | 54.00 [1.00 to 145.00]
  Nef, IL2+, D0 | 1.00 [1.00 to 27.00] | 4.00 [1.00 to 67.00]
  Nef, IL2+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+, D7 | 29.50 [14.50 to 54.50] | 14.00 [1.00 to 81.00]
  Nef, IL2+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+, D14 | 25.00 [14.00 to 56.00] | 14.00 [1.00 to 69.00]
  Nef, IL2+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+, D30 | 1.00 [1.00 to 76.00] | 14.00 [1.00 to 23.00]
  Nef, IL2+, D180 | 21.00 [1.00 to 67.00] | 14.00 [1.00 to 40.00]
  Nef, TNF+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 66.00]
  Nef, TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, TNF+, D7 | 115.00 [16.00 to 155.00] | 97.00 [1.00 to 306.00]
  Nef, TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, TNF+, D14 | 28.00 [1.00 to 135.00] | 95.00 [1.00 to 195.00]
  Nef, TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, TNF+, D30 | 1.00 [1.00 to 22.00] | 10.00 [1.00 to 121.00]
  Nef, TNF+, D180 | 1.00 [1.00 to 20.00] | 1.00 [1.00 to 15.00]
  Nef, IFN+, D0 | 1.00 [1.00 to 23.00] | 1.00 [1.00 to 1.00]
  Nef, IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IFN+, D7 | 14.00 [1.00 to 25.00] | 1.00 [1.00 to 14.00]
  Nef, IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IFN+, D14 | 20.00 [1.00 to 27.00] | 1.00 [1.00 to 23.00]
  Nef, IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 27.00]
  Nef, IFN+, D180 | 14.00 [9.00 to 41.00] | 14.00 [1.00 to 38.00]
  Nef, CD40L+IL2+, D0 | 84.00 [1.00 to 137.00] | 57.00 [28.00 to 165.00]
  Nef, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+, D7 | 199.00 [120.50 to 348.50] | 263.00 [112.00 to 425.00]
  Nef, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+, D14 | 258.00 [57.00 to 424.00] | 191.00 [83.00 to 250.00]
  Nef, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+, D30 | 97.00 [1.00 to 518.00] | 139.00 [82.00 to 230.00]
  Nef, CD40L+IL2+, D180 | 148.00 [94.00 to 243.00] | 129.50 [58.00 to 257.00]
  Nef, CD40L+TNF+, D0 | 3.00 [1.00 to 28.00] | 6.50 [1.00 to 27.00]
  Nef, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+TNF+, D7 | 102.50 [35.00 to 123.00] | 55.00 [42.00 to 137.00]
  Nef, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+TNF+, D14 | 95.00 [11.00 to 162.00] | 56.00 [28.00 to 100.00]
  Nef, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+TNF+, D30 | 56.00 [1.00 to 82.00] | 27.00 [1.00 to 55.00]
  Nef, CD40L+TNF+, D180 | 13.00 [1.00 to 27.00] | 1.00 [1.00 to 27.00]
  Nef, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IFN+, D7 | 14.00 [5.00 to 22.50] | 15.00 [6.00 to 30.00]
  Nef, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IFN+, D14 | 14.00 [1.00 to 19.00] | 1.00 [1.00 to 21.00]
  Nef, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IFN+, D30 | 1.00 [1.00 to 14.00] | 13.00 [1.00 to 25.00]
  Nef, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]

29. Secondary Outcome: Frequency of Antigen (Nef) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Nef, IL2+TNF+, D0 | 9.00 [1.00 to 14.00] | 1.00 [1.00 to 21.00]
  Nef, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+TNF+, D7 | 14.00 [5.50 to 32.50] | 6.00 [1.00 to 42.00]
  Nef, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+TNF+, D14 | 28.00 [1.00 to 56.00] | 14.00 [1.00 to 27.00]
  Nef, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+TNF+, D30 | 1.00 [1.00 to 41.00] | 1.00 [1.00 to 41.00]
  Nef, IL2+TNF+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  Nef, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 11.00]
  Nef, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, TNF+IFN+, D7 | 5.00 [1.00 to 14.50] | 6.00 [1.00 to 20.00]
  Nef, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, TNF+IFN+, D14 | 4.00 [1.00 to 29.00] | 1.00 [1.00 to 22.00]
  Nef, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, TNF+IFN+, D30 | 1.00 [1.00 to 10.00] | 6.00 [1.00 to 27.00]
  Nef, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 7.50 [1.00 to 41.00]
  Nef, CD40L+IL2+TNF+, D0 | 97.00 [81.00 to 167.00] | 93.50 [35.00 to 307.00]
  Nef, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+TNF+, D7 | 268.50 [113.50 to 501.00] | 333.00 [83.00 to 420.00]
  Nef, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+TNF+, D14 | 480.00 [122.00 to 684.00] | 292.00 [139.00 to 555.00]
  Nef, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+TNF+, D30 | 401.00 [72.00 to 627.00] | 191.00 [89.00 to 356.00]
  Nef, CD40L+IL2+TNF+, D180 | 118.00 [103.00 to 175.00] | 107.00 [78.00 to 324.00]
  Nef, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 15.00] | 1.00 [1.00 to 14.00]
  Nef, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+IFN+, D7 | 33.00 [7.50 to 50.50] | 15.00 [8.00 to 49.00]
  Nef, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+IFN+, D14 | 8.00 [1.00 to 56.00] | 10.00 [1.00 to 28.00]
  Nef, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+IFN+, D30 | 14.00 [1.00 to 41.00] | 25.00 [14.00 to 41.00]
  Nef, CD40L+IL2+IFN+, D180 | 14.00 [1.00 to 40.00] | 10.50 [1.00 to 27.00]
  Nef, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+TNF+IFN+, D7 | 12.50 [4.00 to 29.50] | 14.00 [8.00 to 29.00]
  Nef, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40+TNF+IFN+, D14 | 14.00 [1.00 to 26.00] | 10.00 [1.00 to 41.00]
  Nef, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  Nef, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Nef, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 14.00]
  Nef, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  Nef, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  Nef, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  Nef, CD40L+IL2+TNF+IFN+, D0 | 14.00 [1.00 to 31.00] | 12.50 [1.00 to 41.00]
  Nef, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Nef, CD40L+IL2+TNF+IFN+, D7 | 67.50 [28.00 to 109.00] | 80.00 [24.00 to 149.00]
  Nef, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Nef, CD40L+IL2+TNF+IFN+, D14 | 29.00 [14.00 to 80.00] | 28.00 [1.00 to 128.00]
  Nef, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Nef, CD40L+IL2+TNF+IFN+, D30 | 41.00 [1.00 to 95.00] | 38.00 [28.00 to 96.00]
  Nef, CD40L+IL2+TNF+IFN+, D180 | 26.00 [14.00 to 41.00] | 24.00 [1.00 to 75.00]

30. Secondary Outcome: Frequency of Antigen (p17) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P17, CD40L+, D0 | 1.00 [1.00 to 137.00] | 23.50 [1.00 to 103.00]
  P17, CD40L+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+, D7 | 237.50 [1.00 to 405.00] | 217.00 [54.00 to 421.00]
  P17, CD40L+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+, D14 | 112.00 [3.00 to 304.00] | 132.00 [14.00 to 250.00]
  P17, CD40L+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+, D30 | 150.00 [1.00 to 274.00] | 82.00 [1.00 to 236.00]
  P17, CD40L+, D180 | 28.00 [5.00 to 114.00] | 78.50 [60.00 to 108.00]
  P17, IL2+, D0 | 1.00 [1.00 to 28.00] | 1.00 [1.00 to 55.00]
  P17, IL2+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+, D7 | 28.00 [1.00 to 39.00] | 5.00 [1.00 to 47.00]
  P17, IL2+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+, D14 | 8.00 [1.00 to 28.00] | 1.00 [1.00 to 8.00]
  P17, IL2+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+, D30 | 1.00 [1.00 to 1.00] | 14.00 [1.00 to 41.00]
  P17, IL2+, D180 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 24.00]
  P17, TNF+, D0 | 1.00 [1.00 to 89.00] | 1.00 [1.00 to 42.00]
  P17, TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, TNF+, D7 | 40.00 [11.50 to 195.50] | 68.00 [1.00 to 173.00]
  P17, TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, TNF+, D14 | 67.00 [7.00 to 96.00] | 140.00 [14.00 to 184.00]
  P17, TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, TNF+, D30 | 14.00 [1.00 to 41.00] | 82.00 [1.00 to 270.00]
  P17, TNF+, D180 | 1.00 [1.00 to 30.00] | 20.00 [1.00 to 41.00]
  P17, IFN+, D0 | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 27.00]
  P17, IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IFN+, D7 | 1.00 [1.00 to 17.00] | 14.00 [1.00 to 18.00]
  P17, IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IFN+, D14 | 1.00 [1.00 to 8.00] | 9.00 [1.00 to 27.00]
  P17, IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IFN+, D30 | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 14.00]
  P17, IFN+, D180 | 14.00 [1.00 to 19.00] | 1.00 [1.00 to 16.00]
  P17, CD40L+IL2+, D0 | 27.00 [1.00 to 55.00] | 69.00 [1.00 to 124.00]
  P17, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+, D7 | 196.00 [7.00 to 328.50] | 165.00 [56.00 to 380.00]
  P17, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+, D14 | 112.00 [22.00 to 300.00] | 139.00 [109.00 to 340.00]
  P17, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+, D30 | 122.00 [2.00 to 199.00] | 110.00 [58.00 to 248.00]
  P17, CD40L+IL2+, D180 | 138.00 [34.00 to 177.00] | 193.00 [72.00 to 307.00]
  P17, CD40L+TNF+, D0 | 24.00 [1.00 to 43.00] | 1.00 [1.00 to 28.00]
  P17, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+TNF+, D7 | 41.00 [13.00 to 126.50] | 61.00 [27.00 to 99.00]
  P17, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+TNF+, D14 | 28.00 [1.00 to 74.00] | 41.00 [14.00 to 106.00]
  P17, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+TNF+, D30 | 41.00 [16.00 to 83.00] | 14.00 [1.00 to 55.00]
  P17, CD40L+TNF+, D180 | 14.00 [1.00 to 15.00] | 1.00 [1.00 to 19.00]
  P17, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IFN+, D7 | 7.50 [1.00 to 30.50] | 14.00 [1.00 to 37.00]
  P17, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IFN+, D14 | 8.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  P17, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IFN+, D30 | 10.00 [1.00 to 27.00] | 1.00 [1.00 to 27.00]
  P17, CD40L+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]

31. Secondary Outcome: Frequency of Antigen (p17) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P17, IL2+TNF+, D0 | 1.00 [1.00 to 22.00] | 1.00 [1.00 to 14.00]
  P17, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+TNF+, D7 | 1.00 [1.00 to 40.00] | 1.00 [1.00 to 18.00]
  P17, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+TNF+, D14 | 10.00 [1.00 to 25.00] | 1.00 [1.00 to 44.00]
  P17, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+TNF+, D30 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 19.00]
  P17, IL2+TNF+, D180 | 4.00 [1.00 to 27.00] | 1.00 [1.00 to 17.00]
  P17, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, TNF+IFN+, D7 | 7.00 [1.00 to 14.50] | 1.00 [1.00 to 14.00]
  P17, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, TNF+IFN+, D14 | 1.00 [1.00 to 8.00] | 1.00 [1.00 to 14.00]
  P17, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, TNF+IFN+, D30 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 6.00]
  P17, TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+, D0 | 84.00 [26.00 to 97.00] | 115.00 [58.00 to 269.00]
  P17, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+TNF+, D7 | 194.00 [13.00 to 322.00] | 302.00 [27.00 to 824.00]
  P17, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+TNF+, D14 | 192.00 [99.00 to 320.00] | 314.00 [70.00 to 608.00]
  P17, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+TNF+, D30 | 204.00 [37.00 to 947.00] | 203.00 [136.00 to 442.00]
  P17, CD40L+IL2+TNF+, D180 | 94.00 [14.00 to 115.00] | 239.50 [68.00 to 408.00]
  P17, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 15.00] | 1.00 [1.00 to 14.00]
  P17, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+IFN+, D7 | 27.50 [4.00 to 42.00] | 14.00 [1.00 to 49.00]
  P17, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+IFN+, D14 | 1.00 [1.00 to 8.00] | 1.00 [1.00 to 33.00]
  P17, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+IFN+, D30 | 10.00 [1.00 to 14.00] | 14.00 [1.00 to 25.00]
  P17, CD40L+IL2+IFN+, D180 | 13.00 [1.00 to 25.00] | 13.00 [1.00 to 38.00]
  P17, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 10.00]
  P17, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+TNF+IFN+, D7 | 5.00 [1.00 to 21.00] | 14.00 [14.00 to 27.00]
  P17, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40+TNF+IFN+, D14 | 1.00 [1.00 to 14.00] | 11.00 [1.00 to 22.00]
  P17, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  P17, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, IL2+TNF+IFN+, D7 | 4.00 [1.00 to 11.50] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P17, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]
  P17, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 32.00]
  P17, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P17, CD40L+IL2+TNF+IFN+, D7 | 34.50 [5.50 to 129.50] | 31.00 [14.00 to 248.00]
  P17, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P17, CD40L+IL2+TNF+IFN+, D14 | 23.00 [1.00 to 92.00] | 42.00 [1.00 to 155.00]
  P17, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P17, CD40L+IL2+TNF+IFN+, D30 | 40.00 [1.00 to 69.00] | 55.00 [1.00 to 150.00]
  P17, CD40L+IL2+TNF+IFN+, D180 | 14.00 [1.00 to 25.00] | 17.50 [1.00 to 108.00]

32. Secondary Outcome: Frequency of Antigen (p24) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P24, CD40L+, D0 | 79.00 [1.00 to 211.00] | 70.00 [1.00 to 265.00]
  P24, CD40L+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+, D7 | 452.00 [174.00 to 535.50] | 395.00 [80.00 to 477.00]
  P24, CD40L+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+, D14 | 217.00 [76.00 to 359.00] | 154.00 [44.00 to 362.00]
  P24, CD40L+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+, D30 | 86.00 [1.00 to 375.00] | 181.00 [1.00 to 247.00]
  P24, CD40L+, D180 | 118.00 [85.00 to 190.00] | 165.00 [1.00 to 236.00]
  P24, IL2+, D0 | 1.00 [1.00 to 30.00] | 13.00 [1.00 to 72.00]
  P24, IL2+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+, D7 | 40.50 [9.00 to 108.00] | 24.00 [1.00 to 42.00]
  P24, IL2+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+, D14 | 14.00 [7.00 to 29.00] | 5.00 [1.00 to 28.00]
  P24, IL2+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+, D30 | 14.00 [1.00 to 36.00] | 41.00 [14.00 to 73.00]
  P24, IL2+, D180 | 35.00 [14.00 to 68.00] | 2.50 [1.00 to 54.00]
  P24, TNF+, D0 | 1.00 [1.00 to 62.00] | 6.00 [1.00 to 54.00]
  P24, TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, TNF+, D7 | 69.00 [13.00 to 189.00] | 73.00 [1.00 to 245.00]
  P24, TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, TNF+, D14 | 36.00 [1.00 to 138.00] | 53.00 [8.00 to 208.00]
  P24, TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, TNF+, D30 | 1.00 [1.00 to 92.00] | 8.00 [1.00 to 136.00]
  P24, TNF+, D180 | 35.00 [1.00 to 64.00] | 1.00 [1.00 to 13.00]
  P24, IFN+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 29.00]
  P24, IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IFN+, D7 | 4.00 [1.00 to 21.00] | 14.00 [10.00 to 41.00]
  P24, IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IFN+, D14 | 1.00 [1.00 to 12.00] | 14.00 [1.00 to 14.00]
  P24, IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IFN+, D30 | 1.00 [1.00 to 21.00] | 1.00 [1.00 to 11.00]
  P24, IFN+, D180 | 14.00 [1.00 to 65.00] | 1.00 [1.00 to 10.00]
  P24, CD40L+IL2+, D0 | 176.00 [74.00 to 218.00] | 137.00 [1.00 to 323.00]
  P24, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+, D7 | 275.00 [216.50 to 510.50] | 230.00 [140.00 to 658.00]
  P24, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+, D14 | 244.00 [133.00 to 480.00] | 284.00 [57.00 to 430.00]
  P24, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+, D30 | 83.00 [21.00 to 139.00] | 189.00 [149.00 to 329.00]
  P24, CD40L+IL2+, D180 | 234.00 [126.00 to 334.00] | 196.00 [108.00 to 446.00]
  P24, CD40L+TNF+, D0 | 14.00 [1.00 to 26.00] | 21.00 [1.00 to 56.00]
  P24, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+TNF+, D7 | 104.00 [38.50 to 165.50] | 99.00 [41.00 to 160.00]
  P24, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+TNF+, D14 | 86.00 [38.00 to 211.00] | 125.00 [57.00 to 179.00]
  P24, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+TNF+, D30 | 54.00 [17.00 to 113.00] | 42.00 [11.00 to 94.00]
  P24, CD40L+TNF+, D180 | 1.00 [1.00 to 40.00] | 14.50 [1.00 to 27.00]
  P24, CD40L+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 9.00]
  P24, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IFN+, D7 | 12.50 [1.00 to 41.50] | 1.00 [1.00 to 8.00]
  P24, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IFN+, D14 | 11.00 [1.00 to 28.00] | 9.00 [1.00 to 14.00]
  P24, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IFN+, D30 | 1.00 [1.00 to 11.00] | 1.00 [1.00 to 15.00]
  P24, CD40L+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

33. Secondary Outcome: Frequency of Antigen (p24) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 26
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  P24, IL2+TNF+, D0 | 1.00 [1.00 to 9.00] | 1.00 [1.00 to 41.00]
  P24, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+TNF+, D7 | 16.50 [7.00 to 53.50] | 9.00 [1.00 to 42.00]
  P24, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+TNF+, D14 | 27.00 [10.00 to 33.00] | 22.00 [9.00 to 42.00]
  P24, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+TNF+, D30 | 1.00 [1.00 to 60.00] | 14.00 [1.00 to 28.00]
  P24, IL2+TNF+, D180 | 14.00 [1.00 to 24.00] | 27.00 [1.00 to 50.00]
  P24, IL2+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+IFN+, D7 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]
  P24, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, TNF+IFN+, D7 | 7.50 [1.00 to 24.50] | 12.00 [1.00 to 38.00]
  P24, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, TNF+IFN+, D14 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 14.00]
  P24, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, TNF+IFN+, D30 | 1.00 [1.00 to 21.00] | 14.00 [1.00 to 27.00]
  P24, TNF+IFN+, D180 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 17.00]
  P24, CD40L+IL2+TNF+, D0 | 267.00 [145.00 to 314.00] | 135.50 [35.00 to 456.00]
  P24, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+TNF+, D7 | 389.50 [191.00 to 750.00] | 410.00 [277.00 to 678.00]
  P24, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+TNF+, D14 | 569.00 [396.00 to 990.00] | 456.00 [262.00 to 923.00]
  P24, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+TNF+, D30 | 516.00 [49.00 to 692.00] | 379.00 [287.00 to 554.00]
  P24, CD40L+IL2+TNF+, D180 | 233.00 [109.00 to 351.00] | 229.50 [103.00 to 388.00]
  P24, CD40L+IL2+IFN+, D0 | 1.00 [1.00 to 15.00] | 9.50 [1.00 to 27.00]
  P24, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+IFN+, D7 | 20.50 [10.50 to 30.50] | 14.00 [1.00 to 41.00]
  P24, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+IFN+, D14 | 11.00 [1.00 to 47.00] | 23.00 [9.00 to 28.00]
  P24, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+IFN+, D30 | 1.00 [1.00 to 14.00] | 15.00 [9.00 to 41.00]
  P24, CD40L+IL2+IFN+, D180 | 18.00 [1.00 to 42.00] | 14.00 [1.00 to 27.00]
  P24, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+TNF+IFN+, D7 | 12.50 [1.00 to 32.00] | 14.00 [1.00 to 19.00]
  P24, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40+TNF+IFN+, D14 | 14.00 [1.00 to 23.00] | 14.00 [9.00 to 17.00]
  P24, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+TNF+IFN+, D30 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 13.00]
  P24, CD40L+TNF+IFN+, D180 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, IL2+TNF+IFN+, D7 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 6.00]
  P24, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, IL2+TNF+IFN+, D14 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  P24, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 14.00]
  P24, IL2+TNF+IFN+, D180 | 1.00 [1.00 to 22.00] | 1.00 [1.00 to 1.00]
  P24, CD40L+IL2+TNF+IFN+, D0 | 1.00 [1.00 to 44.00] | 14.50 [1.00 to 69.00]
  P24, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  P24, CD40L+IL2+TNF+IFN+, D7 | 140.50 [14.00 to 225.00] | 70.00 [27.00 to 111.00]
  P24, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  P24, CD40L+IL2+TNF+IFN+, D14 | 66.00 [7.00 to 113.00] | 81.00 [32.00 to 114.00]
  P24, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  P24, CD40L+IL2+TNF+IFN+, D30 | 40.00 [13.00 to 83.00] | 57.00 [1.00 to 111.00]
  P24, CD40L+IL2+TNF+IFN+, D180 | 43.00 [26.00 to 52.00] | 22.50 [1.00 to 67.00]

34. Secondary Outcome: Frequency of Antigen (pool_F4co) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: Cytokine/marker co-expression profile was defined as the antigen-specific CD4+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L cytokines as determined by ICS. Determination of F4co was done by stimulating the F4 antigen with a peptide pool spanning (pool_F4co) or by adding individual frequencies of the CD4+ T cell response to each of the 4 antigens (F4co_est).
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Pool_F4co, CD40L+, D0 | 177.00 [1.00 to 280.00] | 264.50 [84.00 to 372.00]
  Pool_F4co, CD40L+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+, D7 | 1809.50 [756.00 to 4021.00] | 2215.00 [991.00 to 2576.00]
  Pool_F4co, CD40L+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+, D14 | 1015.00 [714.00 to 2566.00] | 1175.00 [502.00 to 1520.00]
  Pool_F4co, CD40L+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+, D30 | 653.00 [1.00 to 1250.00] | 650.00 [420.00 to 907.00]
  Pool_F4co, CD40L+, D180 | 497.00 [324.00 to 778.00] | 429.00 [284.00 to 686.00]
  Pool_F4co, IL2+, D0 | 41.00 [5.00 to 66.00] | 57.00 [14.00 to 101.00]
  Pool_F4co, IL2+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+, D7 | 141.50 [48.50 to 245.50] | 81.00 [41.00 to 170.00]
  Pool_F4co, IL2+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+, D14 | 100.00 [14.00 to 190.00] | 92.00 [42.00 to 150.00]
  Pool_F4co, IL2+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+, D30 | 55.00 [20.00 to 105.00] | 97.00 [48.00 to 108.00]
  Pool_F4co, IL2+, D180 | 32.00 [14.00 to 135.00] | 58.50 [35.00 to 108.00]
  Pool_F4co, TNF+, D0 | 20.00 [1.00 to 258.00] | 242.50 [126.00 to 329.00]
  Pool_F4co, TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, TNF+, D7 | 547.50 [310.50 to 687.00] | 625.00 [394.00 to 896.00]
  Pool_F4co, TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, TNF+, D14 | 612.00 [313.00 to 780.00] | 610.00 [386.00 to 977.00]
  Pool_F4co, TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, TNF+, D30 | 225.00 [52.00 to 439.00] | 445.00 [338.00 to 669.00]
  Pool_F4co, TNF+, D180 | 126.00 [76.00 to 148.00] | 56.50 [26.00 to 121.00]
  Pool_F4co, IFN+, D0 | 7.00 [1.00 to 41.00] | 1.00 [1.00 to 20.00]
  Pool_F4co, IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IFN+, D7 | 110.00 [68.50 to 181.50] | 98.00 [27.00 to 135.00]
  Pool_F4co, IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IFN+, D14 | 32.00 [1.00 to 99.00] | 47.00 [18.00 to 129.00]
  Pool_F4co, IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IFN+, D30 | 14.00 [1.00 to 28.00] | 38.00 [8.00 to 56.00]
  Pool_F4co, IFN+, D180 | 35.00 [1.00 to 54.00] | 38.50 [1.00 to 68.00]
  Pool_F4co, CD40L+IL2+, D0 | 469.00 [293.00 to 797.00] | 568.50 [240.00 to 1084.00]
  Pool_F4co, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+, D7 | 1542.50 [899.50 to 2626.00] | 2199.00 [1656.00 to 3507.00]
  Pool_F4co, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+, D14 | 1423.00 [734.00 to 2876.00] | 2037.00 [1276.00 to 2231.00]
  Pool_F4co, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+, D30 | 964.00 [62.00 to 1456.00] | 1277.00 [1019.00 to 1597.00]
  Pool_F4co, CD40L+IL2+, D180 | 961.00 [834.00 to 1369.00] | 1351.50 [976.00 to 1743.00]
  Pool_F4co, CD40L+TNF+, D0 | 102.00 [50.00 to 141.00] | 69.50 [40.00 to 245.00]
  Pool_F4co, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+TNF+, D7 | 514.50 [263.50 to 739.50] | 575.00 [434.00 to 785.00]
  Pool_F4co, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+TNF+, D14 | 706.00 [216.00 to 908.00] | 498.00 [375.00 to 785.00]
  Pool_F4co, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+TNF+, D30 | 399.00 [35.00 to 589.00] | 291.00 [251.00 to 420.00]
  Pool_F4co, CD40L+TNF+, D180 | 81.00 [54.00 to 135.00] | 74.00 [27.00 to 201.00]
  Pool_F4co, CD40L+IFN+, D0 | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 10.00]
  Pool_F4co, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IFN+, D7 | 82.50 [25.00 to 275.50] | 112.00 [39.00 to 152.00]
  Pool_F4co, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IFN+, D14 | 59.00 [27.00 to 85.00] | 56.00 [28.00 to 128.00]
  Pool_F4co, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IFN+, D30 | 21.00 [1.00 to 55.00] | 41.00 [28.00 to 64.00]
  Pool_F4co, CD40L+IFN+, D180 | 14.00 [1.00 to 32.00] | 27.00 [1.00 to 41.00]

35. Secondary Outcome: Frequency of Antigen (pool_F4co) Specific CD4+ T Cells Expressing at Least 2 Markers/Cytokines
Description: as for outcome 34
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  Pool_F4co, IL2+TNF+, D0 | 55.00 [14.00 to 82.00] | 56.00 [12.00 to 141.00]
  Pool_F4co, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+TNF+, D7 | 160.00 [54.00 to 298.50] | 93.00 [42.00 to 149.00]
  Pool_F4co, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+TNF+, D14 | 122.00 [59.00 to 172.00] | 83.00 [57.00 to 224.00]
  Pool_F4co, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+TNF+, D30 | 25.00 [13.00 to 96.00] | 109.00 [82.00 to 127.00]
  Pool_F4co, IL2+TNF+, D180 | 26.00 [14.00 to 108.00] | 59.50 [44.00 to 105.00]
  Pool_F4co, IL2+IFN+, D0 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 1.00]
  Pool_F4co, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+IFN+, D7 | 6.00 [1.00 to 32.00] | 1.00 [1.00 to 25.00]
  Pool_F4co, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+IFN+, D14 | 1.00 [1.00 to 14.00] | 1.00 [1.00 to 20.00]
  Pool_F4co, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+IFN+, D30 | 1.00 [1.00 to 11.00] | 11.00 [1.00 to 14.00]
  Pool_F4co, IL2+IFN+, D180 | 14.00 [1.00 to 16.00] | 14.00 [1.00 to 27.00]
  Pool_F4co, TNF+IFN+, D0 | 1.00 [1.00 to 27.00] | 1.00 [1.00 to 29.00]
  Pool_F4co, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, TNF+IFN+, D7 | 38.00 [18.00 to 106.50] | 56.00 [41.00 to 117.00]
  Pool_F4co, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, TNF+IFN+, D14 | 51.00 [8.00 to 61.00] | 83.00 [42.00 to 97.00]
  Pool_F4co, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, TNF+IFN+, D30 | 27.00 [1.00 to 69.00] | 75.00 [42.00 to 96.00]
  Pool_F4co, TNF+IFN+, D180 | 19.00 [1.00 to 41.00] | 28.00 [1.00 to 54.00]
  Pool_F4co, CD40L+IL2+TNF+, D0 | 792.00 [544.00 to 995.00] | 836.00 [680.00 to 2333.00]
  Pool_F4co, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+TNF+, D7 | 1430.00 [961.00 to 3040.00] | 2764.00 [1649.00 to 3631.00]
  Pool_F4co, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+TNF+, D14 | 2032.00 [1164.00 to 3906.00] | 2804.00 [2313.00 to 3500.00]
  Pool_F4co, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+TNF+, D30 | 2243.00 [215.00 to 3151.00] | 2137.00 [1764.00 to 2653.00]
  Pool_F4co, CD40L+IL2+TNF+, D180 | 1146.00 [682.00 to 1481.00] | 1246.00 [945.00 to 2046.00]
  Pool_F4co, CD40L+IL2+IFN+, D0 | 28.00 [14.00 to 44.00] | 30.50 [1.00 to 96.00]
  Pool_F4co, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+IFN+, D7 | 140.00 [83.00 to 426.00] | 204.00 [84.00 to 294.00]
  Pool_F4co, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+IFN+, D14 | 96.00 [55.00 to 221.00] | 151.00 [119.00 to 245.00]
  Pool_F4co, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+IFN+, D30 | 24.00 [1.00 to 179.00] | 109.00 [58.00 to 154.00]
  Pool_F4co, CD40L+IL2+IFN+, D180 | 116.00 [27.00 to 188.00] | 60.50 [29.00 to 176.00]
  Pool_F4co, CD40L+TNF+IFN+, D0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 12.00]
  Pool_F4co, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+TNF+IFN+, D7 | 70.00 [27.50 to 155.00] | 97.00 [15.00 to 168.00]
  Pool_F4co, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40+TNF+IFN+, D14 | 74.00 [27.00 to 141.00] | 85.00 [42.00 to 163.00]
  Pool_F4co, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+TNF+IFN+, D30 | 55.00 [1.00 to 122.00] | 82.00 [31.00 to 127.00]
  Pool_F4co, CD40L+TNF+IFN+, D180 | 27.00 [13.00 to 41.00] | 27.00 [14.00 to 43.00]
  Pool_F4co, IL2+TNF+IFN+, D0 | 1.00 [1.00 to 14.00] | 11.00 [1.00 to 14.00]
  Pool_F4co, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, IL2+TNF+IFN+, D7 | 18.50 [4.50 to 68.00] | 14.00 [1.00 to 41.00]
  Pool_F4co, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, IL2+TNF+IFN+, D14 | 8.00 [1.00 to 17.00] | 14.00 [1.00 to 28.00]
  Pool_F4co, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, IL2+TNF+IFN+, D30 | 1.00 [1.00 to 22.00] | 17.00 [13.00 to 27.00]
  Pool_F4co, IL2+TNF+IFN+, D180 | 13.00 [1.00 to 14.00] | 17.50 [1.00 to 40.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D0 | 95.00 [44.00 to 206.00] | 147.00 [1.00 to 304.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D7 | 285.50 [152.00 to 798.50] | 484.00 [226.00 to 926.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D14 | 337.00 [176.00 to 802.00] | 639.00 [304.00 to 922.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  Pool_F4co, CD40L+IL2+TNF+IFN+, D30 | 244.00 [1.00 to 537.00] | 413.00 [183.00 to 757.00]
  Pool_F4co, CD40L+IL2+TNF+IFN+, D180 | 163.00 [80.00 to 438.00] | 216.00 [121.00 to 407.00]

36. Secondary Outcome: Frequency of Antigen (F4co_est) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 34
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  F4co_est, CD40L+, D0 | 562.00 [166.00 to 932.00] | 270.50 [101.00 to 828.00]
  F4co_est, CD40L+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+, D7 | 2050.50 [1173.50 to 5806.00] | 2296.00 [1038.00 to 2839.00]
  F4co_est, CD40L+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+, D14 | 1106.00 [411.00 to 2472.00] | 1108.00 [404.00 to 1713.00]
  F4co_est, CD40L+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+, D30 | 584.00 [4.00 to 1965.00] | 697.00 [517.00 to 959.00]
  F4co_est, CD40L+, D180 | 543.00 [442.00 to 730.00] | 507.00 [349.00 to 895.00]
  F4co_est, IL2+, D0 | 54.00 [29.00 to 105.00] | 138.00 [30.00 to 235.00]
  F4co_est, IL2+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+, D7 | 201.50 [108.50 to 386.00] | 165.00 [58.00 to 175.00]
  F4co_est, IL2+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+, D14 | 130.00 [96.00 to 263.00] | 92.00 [30.00 to 152.00]
  F4co_est, IL2+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+, D30 | 75.00 [4.00 to 206.00] | 134.00 [70.00 to 180.00]
  F4co_est, IL2+, D180 | 82.00 [44.00 to 294.00] | 93.00 [63.00 to 191.00]
  F4co_est, TNF+, D0 | 192.00 [69.00 to 235.00] | 129.50 [67.00 to 488.00]
  F4co_est, TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, TNF+, D7 | 844.00 [272.50 to 1066.50] | 635.00 [297.00 to 1151.00]
  F4co_est, TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, TNF+, D14 | 388.00 [267.00 to 605.00] | 477.00 [314.00 to 1023.00]
  F4co_est, TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, TNF+, D30 | 194.00 [66.00 to 300.00] | 608.00 [194.00 to 654.00]
  F4co_est, TNF+, D180 | 191.00 [19.00 to 243.00] | 40.50 [4.00 to 123.00]
  F4co_est, IFN+, D0 | 43.00 [11.00 to 71.00] | 42.00 [14.00 to 58.00]
  F4co_est, IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IFN+, D7 | 141.50 [44.50 to 189.50] | 93.00 [32.00 to 150.00]
  F4co_est, IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IFN+, D14 | 30.00 [17.00 to 102.00] | 71.00 [17.00 to 112.00]
  F4co_est, IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IFN+, D30 | 24.00 [4.00 to 57.00] | 30.00 [4.00 to 71.00]
  F4co_est, IFN+, D180 | 120.00 [45.00 to 139.00] | 36.50 [4.00 to 87.00]
  F4co_est, CD40L+IL2+, D0 | 659.00 [467.00 to 722.00] | 761.50 [231.00 to 1073.00]
  F4co_est, CD40L+IL2+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+, D7 | 2048.00 [1017.50 to 2779.50] | 2496.00 [1282.00 to 3250.00]
  F4co_est, CD40L+IL2+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+, D14 | 1724.00 [802.00 to 3005.00] | 1860.00 [1493.00 to 2091.00]
  F4co_est, CD40L+IL2+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+, D30 | 1042.00 [98.00 to 1472.00] | 1217.00 [1129.00 to 1643.00]
  F4co_est, CD40L+IL2+, D180 | 1184.00 [883.00 to 1732.00] | 1309.50 [876.00 to 1721.00]
  F4co_est, CD40L+TNF+, D0 | 74.00 [56.00 to 177.00] | 95.00 [46.00 to 174.00]
  F4co_est, CD40L+TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+TNF+, D7 | 491.50 [233.00 to 907.00] | 591.00 [326.00 to 721.00]
  F4co_est, CD40L+TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+TNF+, D14 | 554.00 [246.00 to 747.00] | 596.00 [306.00 to 864.00]
  F4co_est, CD40L+TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+TNF+, D30 | 382.00 [87.00 to 593.00] | 234.00 [210.00 to 288.00]
  F4co_est, CD40L+TNF+, D180 | 109.00 [59.00 to 128.00] | 63.50 [49.00 to 146.00]
  F4co_est, CD40L+IFN+, D0 | 4.00 [4.00 to 15.00] | 9.00 [4.00 to 17.00]
  F4co_est, CD40L+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IFN+, D7 | 123.50 [38 to 254.50] | 127.00 [32.00 to 197.00]
  F4co_est, CD40L+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IFN+, D14 | 68.00 [33.00 to 122.00] | 60.00 [43.00 to 87.00]
  F4co_est, CD40L+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IFN+, D30 | 24.00 [4.00 to 75.00] | 61.00 [30.00 to 84.00]
  F4co_est, CD40L+IFN+, D180 | 17.00 [4.00 to 35.00] | 30.00 [17.00 to 45.00]

37. Secondary Outcome: Frequency of Antigen (F4co_est) Specific CD4+ T Cells Expressing at Least 2 Markers/ Cytokines
Description: as for outcome 34
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
T cells/million cells
  F4co_est, IL2+TNF+, D0 | 37.00 [24.00 to 117.00] | 34.50 [4.00 to 178.00]
  F4co_est, IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+TNF+, D7 | 165.00 [69.50 to 267.00] | 86.00 [66.00 to 110.00]
  F4co_est, IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+TNF+, D14 | 103.00 [56.00 to 284.00] | 49.00 [43.00 to 210.00]
  F4co_est, IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+TNF+, D30 | 30.00 [21.00 to 192.00] | 82.00 [31.00 to 175.00]
  F4co_est, IL2+TNF+, D180 | 43.00 [28.00 to 123.00] | 87.50 [70.00 to 187.00]
  F4co_est, IL2+IFN+, D0 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  F4co_est, IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+IFN+, D7 | 17.00 [4.00 to 43.50] | 12.00 [4.00 to 18.00]
  F4co_est, IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+IFN+, D14 | 10.00 [4.00 to 31.00] | 4.00 [4.00 to 17.00]
  F4co_est, IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+IFN+, D30 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 18.00]
  F4co_est, IL2+IFN+, D180 | 4.00 [4.00 to 30.00] | 17.00 [4.00 to 30.00]
  F4co_est, TNF+IFN+, D0 | 17.00 [4.00 to 32.00] | 14.00 [4.00 to 18.00]
  F4co_est, TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, TNF+IFN+, D7 | 45.00 [29.00 to 116.50] | 72.00 [30.00 to 88.00]
  F4co_est, TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, TNF+IFN+, D14 | 56.00 [4.00 to 83.00] | 64.00 [18.00 to 71.00]
  F4co_est, TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, TNF+IFN+, D30 | 35.00 [21.00 to 57.00] | 86.00 [36.00 to 100.00]
  F4co_est, TNF+IFN+, D180 | 17.00 [4.00 to 31.00] | 59.50 [17.00 to 96.00]
  F4co_est, CD40L+IL2+TNF+, D0 | 1050.00 [566.00 to 1215.00] | 972.50 [398.00 to 2654.00]
  F4co_est, CD40L+IL2+TNF+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+TNF+, D7 | 1587.00 [1067.50 to 3516.50] | 3392.00 [1962.00 to 4350.00]
  F4co_est, CD40L+IL2+TNF+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+TNF+, D14 | 2652.00 [1588.00 to 4691.00] | 3279.00 [2871.00 to 4311.00]
  F4co_est, CD40L+IL2+TNF+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+TNF+, D30 | 2635.00 [202.00 to 3943.00] | 2593.00 [1885.00 to 2825.00]
  F4co_est, CD40L+IL2+TNF+, D180 | 1088.00 [584.00 to 1552.00] | 1288.50 [984.00 to 2408.00]
  F4co_est, CD40L+IL2+IFN+, D0 | 51.00 [26.00 to 96.00] | 45.00 [29.00 to 82.00]
  F4co_est, CD40L+IL2+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+IFN+, D7 | 158.50 [77.50 to 429.00] | 254.00 [118.00 to 327.00]
  F4co_est, CD40L+IL2+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+IFN+, D14 | 107.00 [57.00 to 226.00] | 157.00 [99.00 to 212.00]
  F4co_est, CD40L+IL2+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+IFN+, D30 | 46.00 [4.00 to 153.00] | 139.00 [97.00 to 182.00]
  F4co_est, CD40L+IL2+IFN+, D180 | 123.00 [70.00 to 176.00] | 104.00 [30.00 to 190.00]
  F4co_est, CD40L+TNF+IFN+, D0 | 4.00 [4.00 to 17.00] | 8.50 [4.00 to 26.00]
  F4co_est, CD40L+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+TNF+IFN+, D7 | 86.50 [64.00 to 144.00] | 111.00 [48.00 to 168.00]
  F4co_est, CD40+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40+TNF+IFN+, D14 | 82.00 [43.00 to 142.00] | 85.00 [31.00 to 154.00]
  F4co_est, CD40L+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+TNF+IFN+, D30 | 43.00 [12.00 to 99.00] | 44.00 [32.00 to 74.00]
  F4co_est, CD40L+TNF+IFN+, D180 | 16.00 [4.00 to 19.00] | 22.50 [4.00 to 43.00]
  F4co_est, IL2+TNF+IFN+, D0 | 4.00 [4.00 to 15.00] | 4.00 [4.00 to 17.00]
  F4co_est, IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, IL2+TNF+IFN+, D7 | 21.00 [16.00 to 35.00] | 30.00 [11.00 to 58.00]
  F4co_est, IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, IL2+TNF+IFN+, D14 | 17.00 [4.00 to 30.00] | 17.00 [4.00 to 57.00]
  F4co_est, IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, IL2+TNF+IFN+, D30 | 4.00 [4.00 to 14.00] | 27.00 [17.00 to 43.00]
  F4co_est, IL2+TNF+IFN+, D180 | 25.00 [17.00 to 69.00] | 30.00 [4.00 to 34.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D0 | 107.00 [71.00 to 142.00] | 138.00 [44.00 to 207.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D7: number analyzed (Participants) | 12 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D7 | 348.00 [246.50 to 1074.50] | 512.00 [235.00 to 1098.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D14: number analyzed (Participants) | 13 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D14 | 457.00 [97.00 to 608.00] | 601.00 [250.00 to 938.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D30: number analyzed (Participants) | 11 | 13
  F4co_est, CD40L+IL2+TNF+IFN+, D30 | 284.00 [21.00 to 747.00] | 384.00 [206.00 to 854.00]
  F4co_est, CD40L+IL2+TNF+IFN+, D180 | 134.00 [97.00 to 367.00] | 244.00 [82.00 to 419.00]

38. Secondary Outcome: Anti- RT, Nef, p17, p24 and F4co Antibody Concentrations
Description: Antibody concentrations were expressed as geometric mean concentrations (GMCs), given in milli-enzyme-linked immunosorbent assay (ELISA) units per millilitre (mEL.U/mL).
Time Frame: At Day 0, 7, 14, 30 and 180
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mEL.U/mL
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Number analyzed (Participants) | 13 | 14
mEL.U/mL
  Anti-RT, Day 0 | 154.0 [95.8 to 247.5] | 198.4 [99.0 to 397.7]
  Anti-RT, Day 7 | 31465.3 [13461.3 to 73549.0] | 39928.9 [21751.5 to 73297.1]
  Anti-RT, Day 14 | 79774.0 [50733.0 to 125439.0] | 59932.0 [37464.8 to 95872.6]
  Anti-RT, Day 30 | 71028.8 [48687.2 to 103622.7] | 57653.6 [35758.1 to 92956.1]
  Anti-RT, Day 180 | 27286.9 [18489.9 to 40269.3] | 26520.6 [14387.7 to 48885.0]
  Anti-Nef, Day 0 | 394.6 [243.4 to 639.5] | 536.3 [251.9 to 1141.7]
  Anti-Nef, Day 7 | 38430.3 [15157.6 to 97435.4] | 38621.8 [19829.5 to 75223.5]
  Anti-Nef, Day 14 | 113387.2 [62469.0 to 205808.7] | 63283.3 [36141.0 to 110809.8]
  Anti-Nef, Day 30 | 77192.3 [39847.3 to 149537.1] | 42709.2 [21389.9 to 85277.2]
  Anti-Nef, Day 180 | 25141.1 [14744.0 to 42870.2] | 21371.8 [10260.3 to 44517.0]
  Anti-p17, Day 0 | 93.5 [93.5 to 93.5] | 98.9 [87.6 to 111.6]
  Anti-p17, Day 7 | 1599.4 [704.7 to 3629.7] | 1121.5 [390.5 to 3220.5]
  Anti-p17, Day 14 | 5069.8 [2356.8 to 10906.1] | 1763.3 [545.6 to 5699.3]
  Anti-p17, Day 30 | 5148.5 [2493.1 to 10632.1] | 1610.1 [436.1 to 5944.5]
  Anti-p17, Day 180 | 1115.5 [498.9 to 2493.9] | 639.0 [215.1 to 1899.0]
  Anti-p24, Day 0 | 377.4 [271.1 to 525.3] | 483.3 [222.0 to 1051.9]
  Anti-p24, Day 7 | 31533.9 [14691.0 to 67686.9] | 36200.9 [22284.8 to 58807.3]
  Anti-p24, Day 14 | 78313.7 [51412.0 to 119292.0] | 59655.5 [40848.9 to 87120.6]
  Anti-p24, Day 30 | 61372.0 [41678.5 to 90370.9] | 49619.3 [31879.0 to 77231.9]
  Anti-p24, Day 180 | 27590.9 [18812.2 to 40466.2] | 27545.3 [16128.6 to 47043.3]
  Anti-F4co, Day 0 | 217.8 [147.1 to 322.3] | 330.2 [194.0 to 562.0]
  Anti-F4co, Day 7 | 37905.7 [16622.6 to 86438.8] | 39948.9 [24778.8 to 64406.3]
  Anti-F4co, Day 14 | 83863.4 [56912.6 to 123576.8] | 63951.9 [45830.2 to 89239.0]
  Anti-F4co, Day 30 | 74791.3 [50872.9 to 109955.1] | 65633.5 [42838.2 to 100558.8]
  Anti-F4co, Day 180 | 42847.4 [28001.7 to 65563.8] | 40715.4 [24865.2 to 66669.5]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7 Day (Day 0 to Day 6) post-vaccination period; Unsolicited AEs until Day 29 post-vaccination; SAEs during the entire study period (from Day 0 up to Day 360).
Arm/Group | GSK732461+Nivaquine Group | GSK732461 Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 13/13 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK732461+Nivaquine Group (N=13) | GSK732461 Group (N=15)
Chills (General disorders) | 1 | 6
Hangover (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 2
Injection site haemorrhage (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 — 1 subject in the GSK732461+Nivaquine group reported gastroenteritis 1 day before vaccination
Rhinitis (Infections and infestations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 9 | 14
Gastro-intestinal symptoms (General disorders) | 6 | 5
Headache (General disorders) | 9 | 13
Temperature (Orally) (General disorders) | 8 | 10
Pain (General disorders) | 13 | 14
Redness (General disorders) | 3 | 6
Swelling (General disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.